CLINICAL TRIAL: NCT02804763
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study Followed by an Observational Period to Evaluate the Efficacy and Safety of Dapirolizumab Pegol in Subjects With Moderately to Severely Active Systemic Lupus Erythematosus
Brief Title: A Phase 2 Efficacy and Safety Study of Dapirolizumab Pegol (DZP) in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL0023; 2015-004457-40 (EudraCT Number)
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic Lupus Erythematosus (SLE); Dapirolizumab Pegol (DZP)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — dapirolizumab pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo in a specified sequence for a total of 24 weeks
  Interventions: Drug: Placebo
- DZP dose 1 (Experimental): Dapirolizumab pegol (DZP) dose 1 in a specified sequence for a total of 24 weeks
  Interventions: Drug: Dapirolizumab pegol (DZP)
- DZP dose 2 (Experimental): Dapirolizumab pegol (DZP) dose 2 in a specified sequence for a total of 24 weeks
  Interventions: Drug: Dapirolizumab pegol (DZP)
- DZP dose 3 (Experimental): Dapirolizumab pegol (DZP) dose 3 in a specified sequence for a total of 24 weeks
  Interventions: Drug: Dapirolizumab pegol (DZP)

INTERVENTIONS:
Drug: Placebo — Solution for infusion, 0,9% saline
  Arms: Placebo
Drug: Dapirolizumab pegol (DZP) — Solution for infusion
  Arms: DZP dose 1; DZP dose 2; DZP dose 3

SUMMARY:
The purpose is to evaluate the efficacy and safety of three different doses of Dapirolizumab Pegol (DZP) versus placebo in adult subjects with moderately to severely active systemic Lupus Erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Systemic Lupus Erythematosus (SLE) confirmed by Systemic Lupus International Collaborating Clinics (SLICC) classification criteria
* Moderate to severe SLE disease activity
* Evidence for at least 1 of the following SLE markers:

  * Anti-dsDNA antibodies confirmed by central laboratory or
  * Low complement confirmed by central laboratory or
  * Antinuclear antibody (ANA) titer of >= 1:80 in combination with at least 1 of the following: Historical positivity for anti-dsDNA or Positivity for extractable nuclear antigen (anti-ENA) confirmed by central laboratory
* The subject is receiving stable SLE standard-of-care medication

Exclusion Criteria:

* Mixed connective tissue disease, scleroderma, and/or overlap syndromes of SLE
* Subjects with severe neuropsychiatric SLE or other neurological symptoms that in the opinion of the Investigator, would prevent the subject from completing protocol required procedures and assessments.
* New or worsening Class III or IV lupus nephritis
* Chronic kidney failure stage 3b
* Evidence of human immunodeficiency virus (HIV) infection, agammaglobulinemias, T-cell deficiencies, or human T-cell lymphotropic virus-1 infection at any time prior to or during the study
* Clinically significant active or latent infection (eg. chronic viral hepatitis B or C)
* Known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent TB (LTB) infection
* Live/live attenuated vaccines within 6 weeks prior to the first study drug infusion (Visit 2) or who plan to receive these vaccines during the study or 12 weeks after the final dose of study drug
* History of thromboembolic events within 12 months of screening
* Subject has used protocol defined prohibited medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (71):
- United States (25):
  - Sl0023 312, Birmingham, Alabama
  - Sl0023 307, El Cajon, California
  - Sl0023 309, El Cajon, California
  - Sl0023 323, Huntington Beach, California
  - Sl0023 311, Los Angeles, California
  - Sl0023 314, Thousand Oaks, California
  - Sl0023 302, Upland, California
  - Sl0023 326, New Haven, Connecticut
  - Sl0023 304, Clearwater, Florida
  - Sl0023 322, DeBary, Florida
  - Sl0023 321, Miami, Florida
  - Sl0023 301, Miami Lakes, Florida
  - Sl0023 319, Palm Harbor, Florida
  - Sl0023 310, Tampa, Florida
  - Sl0023 324, Atlanta, Georgia
  - Sl0023 327, Stockbridge, Georgia
  - Sl0023 320, Idaho Falls, Idaho
  - Sl0023 306, Albuquerque, New Mexico
  - Sl0023 313, Lake Success, New York
  - Sl0023 305, Oklahoma City, Oklahoma
  - Sl0023 315, Jackson, Tennessee
  - Sl0023 308, Memphis, Tennessee
  - Sl0023 317, Amarillo, Texas
  - Sl0023 303, Houston, Texas
  - Sl0023 328, Spokane, Washington
- Bulgaria (2):
  - Sl0023 101, Plovdiv
  - Sl0023 102, Plovdiv
- Chile (4):
  - Sl0023 202, Providencia
  - Sl0023 203, Providencia
  - Sl0023 201, Puerto Varas
  - Sl0023 204, Viña del Mar
- Colombia (6):
  - Sl0023 213, Barranquilla
  - Sl0023 212, Bogotá
  - Sl0023 214, Bogotá
  - Sl0023 216, Bucaramanga
  - Sl0023 211, Chía
  - Sl0023 215, Medellín
- Germany (2):
  - Sl0023 341, Hanover
  - Sl0023 113, Leipzig
- Sl0023 124, Debrecen, Hungary
- Mexico (4):
  - Sl0023 225, Guadalajara
  - Sl0023 224, León
  - Sl0023 221, México
  - Sl0023 222, San Luis Potosí City
- Peru (4):
  - Sl0023 232, Arequipa
  - Sl0023 231, Lima
  - Sl0023 234, Lima
  - Sl0023 235, Lima
- Poland (6):
  - Sl0023 133, Bytom
  - Sl0023 138, Lodz
  - Sl0023 136, Lublin
  - Sl0023 131, Poznan
  - Sl0023 134, Sosnowiec
  - Sl0023 135, Warsaw
- Romania (4):
  - Sl0023 146, Brasov
  - Sl0023 142, Bucharest
  - Sl0023 144, Cluj-Napoca
  - Sl0023 141, Galati
- Russia (6):
  - Sl0023 157, Kazan'
  - Sl0023 156, Kemerovo
  - Sl0023 152, Saint Petersburg
  - Sl0023 155, Voronezh
  - Sl0023 151, Yaroslavl
  - Sl0023 153, Yekaterinburg
- Spain (3):
  - Sl0023 161, Barcelona
  - Sl0023 162, Madrid
  - Sl0023 166, Santa Cruz de Tenerife
- Ukraine (4):
  - Sl0023 172, Kyiv
  - Sl0023 175, Kyiv
  - Sl0023 171, Odesa
  - Sl0023 173, Vinnytsia

REFERENCES:
- [Derived] Acharya C, Magnusson MO, Vajjah P, Oliver R, Zamacona M. Population Pharmacokinetics and Exposure-Response for Dapirolizumab Pegol From a Phase 2b Trial in Patients With Systemic Lupus Erythematosus. J Clin Pharmacol. 2023 Apr;63(4):435-444. doi: 10.1002/jcph.2188. Epub 2023 Jan 9. PMID 36453450
- [Derived] Morel T, Cano S, Bartlett SJ, Gordon C, Haier B, Regnault A, Schneider M, Stach C, Cleanthous S. The FATIGUE-PRO: a new patient-reported outcome instrument to quantify fatigue in patients affected by systemic lupus erythematosus. Rheumatology (Oxford). 2022 Aug 3;61(8):3329-3340. doi: 10.1093/rheumatology/keab920. PMID 34897375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in June 2016 and concluded in November 2018.
Pre-assignment Details: The study included a 4-week Screening Period, a 24-week Double-Blind Treatment Period and a 24-week Observational Period.
  Participant Flow refers to the Randomized Set.
Groups:
- SOC + Placebo iv Q4W: This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive Placebo intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period.
- SOC + DZP 6mg/kg iv Q4W: This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 6 milligrams (mg)/kilogram (kg) intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period.
- SOC + DZP 24mg/kg iv Q4W: This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 24mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period.
- SOC + DZP 45mg/kg iv Q4W: This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 45mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period.
Period: Double-Blind Period (Week 1 to Week 24)
Arm/Group | SOC + Placebo iv Q4W | SOC + DZP 6mg/kg iv Q4W | SOC + DZP 24mg/kg iv Q4W | SOC + DZP 45mg/kg iv Q4W
Started | 45 | 45 | 45 | 47
Completed Week 24 | 44 | 45 | 44 | 45
Finished Wk24 Began Observational Period | 44 | 44 | 44 | 45
Completed | 44 | 44 | 44 | 45
Not Completed | 1 | 1 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Consent withdrawal after Week 24 | 0 | 1 | 0 | 0
Period: Observational Period (Wk 24 to Wk 48)
Arm/Group | SOC + Placebo iv Q4W | SOC + DZP 6mg/kg iv Q4W | SOC + DZP 24mg/kg iv Q4W | SOC + DZP 45mg/kg iv Q4W
Started | 44 | 44 | 44 | 45
Completed | 38 | 43 | 41 | 42
Not Completed | 6 | 1 | 3 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 2 | 2
Not completed — Patient moved out of state | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all study participants who were randomized and received at least 1 dose (any amount) of study drug.
Arm/Group | SOC + Placebo iv Q4W | SOC + DZP 6mg/kg iv Q4W | SOC + DZP 24mg/kg iv Q4W | SOC + DZP 45mg/kg iv Q4W | Total Title
Number analyzed (Participants) | 45 | 45 | 45 | 47 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 44 | 46 | 178
  >=65 years | 1 | 1 | 1 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.50 (12.79) | 40.81 (11.55) | 42.77 (10.42) | 38.94 (12.92) | 41.48 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 40 | 43 | 166
  Male | 4 | 3 | 5 | 4 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 1 | 5
  Asian | 1 | 0 | 1 | 0 | 2
  Black | 1 | 4 | 1 | 6 | 12
  White | 27 | 26 | 33 | 27 | 113
  Other/Mixed | 14 | 14 | 9 | 13 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004)-Based Composite Lupus Assessment (BICLA) (mNRI) Response Across 3 Doses of Dapirolizumab Pegol (DZP) and Placebo (PBO) at Week 24
Description: The primary efficacy variable was assessed by establishing if there was a dose response relationship between BICLA response at Week 24 and dose, using Multiple Comparison Procedure - Modelling (MCP-Mod). Four candidate dose-response models were evaluated: a linear model, a logistic model, and 2 Emax models, and the MCP-Mod methodology controlled for multiplicity.
  BICLA response was defined as meeting all of the following criteria:
  1. BILAG 2004 improvement: A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤ 1 new B.
  2. No worsening in Systemic Lupus Erythematosus Activity Index 2000 (SLEDAI-2K), defined as no increase in SLEDAI-2K total score.
  3. No worsening in Physician's Global Assessment of Disease Activity (PGA), defined as < 10 millimeter (mm) increase on a 100 mm visual analog scale (VAS).
  4. No disallowed changes in concomitant medications, mainly including increases in corticosteroids, immunosuppressants, and antimalarials.
Time Frame: Week 24
Population: The Full Analysis Set (FAS) consisted of all participants in the Randomized Set with the exception of 1 study participant who received less than 1 full dose during the study and 5 study participants who were randomized at Site 321.
  Missing values were imputed using a modified non-responder imputation (mNRI).
Measure: Number; unit: percentage of participants
Groups:
- SOC + Placebo iv Q4W (FAS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive Placebo intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the Full Analysis Set (FAS).
- SOC + DZP 6mg/kg iv Q4W (FAS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 6mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the FAS.
- SOC + DZP 24mg/kg iv Q4W (FAS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 24mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the FAS.
- SOC + DZP 45mg/kg iv Q4W (FAS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 45mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the FAS.
Arm/Group | SOC + Placebo iv Q4W (FAS) | SOC + DZP 6mg/kg iv Q4W (FAS) | SOC + DZP 24mg/kg iv Q4W (FAS) | SOC + DZP 45mg/kg iv Q4W (FAS)
Number analyzed (Participants) | 43 | 43 | 44 | 46
percentage of participants | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 6mg/kg iv Q4W (FAS) vs SOC + DZP 24mg/kg iv Q4W (FAS) vs SOC + DZP 45mg/kg iv Q4W (FAS); Multiple contrast testing (MCP-mod methodology) was used to test for a statistically significant dose-response relationship between the primary endpoint (BICLA at Week 24) and dose, which would indicate a drug effect of DZP over Placebo. The best fitting statistically significant model could be used to estimate the dose needed to achieve desired treatment effect; Test type: Superiority; p = 0.0727, MCP-Mod — The lowest p-value (z-statistic with the highest value) was used to establish proof of dose response

2. Secondary Outcome: The Percentage of Participants With BICLA (mNRI) Response in the Individual Dose Groups at Week 24
Description: BICLA response was defined as meeting all of the following criteria:
  1. BILAG 2004 improvement: A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤ 1 new B.
  2. No worsening in Systemic Lupus Erythematosus Activity Index 2000 (SLEDAI-2K), defined as no increase in SLEDAI-2K total score.
  3. No worsening in Physician's Global Assessment of Disease Activity (PGA), defined as < 10 millimeter (mm) increase on a 100 mm visual analog scale (VAS).
  4. No disallowed changes in concomitant medications, mainly including increases in corticosteroids, immunosuppressants, and antimalarials.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SOC + Placebo iv Q4W (FAS) | SOC + DZP 6mg/kg iv Q4W (FAS) | SOC + DZP 24mg/kg iv Q4W (FAS) | SOC + DZP 45mg/kg iv Q4W (FAS)
Number analyzed (Participants) | 43 | 43 | 44 | 46
percentage of participants | 37.2 | 48.8 | 54.5 | 52.2
Statistical Analysis 1: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 6mg/kg iv Q4W (FAS); Missing values were imputed using modified non-responder imputation (mNRI) dataset: at most 1 missing BICLA (mNRI) component (scale) may have been carried forward from the immediately preceding visit, and missing data in the individual items within scales may have been carried forward from the immediately preceding visit. If there was still missing data after this limited imputation, the study participant was counted as a non-responder on the BICLA (mNRI) for that visit; Test type: Superiority; p = 0.2699, Chi-squared — Generalized linear models with factors for treatment and corticosteroid strata were fit using a logit link function for the odds ratios and p-values; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.7 to 3.8]
Statistical Analysis 2: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 24mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1036, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.0, 95% CI 2-sided [0.9 to 4.8]
Statistical Analysis 3: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 45mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1518, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.9, 95% CI 2-sided [0.8 to 4.3]
Statistical Analysis 4: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 6mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Chi-squared — Crude difference in proportion responding and standard Wald asymptotic 95 % CI based on the normal approximation to the binomial distribution; Difference vs PBO = 11.6, 95% CI 2-sided [-9.2 to 32.4] — Difference and 95 % Wald CI in proportion of responders for SOC + DZP dose 1 iv Q4W (FAS) versus SOC + Placebo iv Q4W (FAS)
Statistical Analysis 5: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 24mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Chi-squared — [p-value comment as in outcome 2, analysis 4]; Difference vs PBO = 17.3, 95% CI 2-sided [-3.3 to 38.0] — Difference and 95 % Wald CI in proportion of responders for SOC + DZP dose 2 iv Q4W (FAS) versus SOC + Placebo iv Q4W (FAS)
Statistical Analysis 6: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 45mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Chi-squared — [p-value comment as in outcome 2, analysis 4]; Difference vs PBO = 15.0, 95% CI 2-sided [-5.5 to 35.4] — Difference and 95 % Wald CI in proportion of responders for SOC + DZP dose 3 iv Q4W (FAS) versus SOC + Placebo iv Q4W (FAS)
Statistical Analysis 7: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 6mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Chi-squared — Generalized linear models with factors for treatment and corticosteroid strata were fit using an identity link function for the LS mean differences; LS Mean Difference vs PBO = 11.9, 95% CI 2-sided [-8.7 to 32.5]
Statistical Analysis 8: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 24mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Chi-squared — [p-value comment as in outcome 2, analysis 7]; LS Mean Difference vs PBO = 17.6, 95% CI 2-sided [-3.2 to 38.3]
Statistical Analysis 9: Comparison: SOC + Placebo iv Q4W (FAS) vs SOC + DZP 45mg/kg iv Q4W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Chi-squared — [p-value comment as in outcome 2, analysis 7]; LS Mean Difference vs PBO = 15.2, 95% CI 2-sided [-5.2 to 35.6]

3. Secondary Outcome: Percentage of Participants With at Least One Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An adverse event (AE) was therefore any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. All AEs that occurred during the study were considered related unless clearly unrelated.
Time Frame: From Baseline (Week 1) until end of the study (Week 48)
Population: The Safety Set (SS) consisted of all study participants who were randomized and received at least 1 dose (any amount) of study drug.
Measure: Number; unit: percentage of participants
Groups:
- SOC + Placebo iv Q4W (SS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive Placebo intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the Safety Set (SS).
- SOC + DZP 6mg/kg iv Q4W (SS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 6mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the SS.
- SOC + DZP 24mg/kg iv Q4W (SS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 24mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the SS.
- SOC + DZP 45mg/kg iv Q4W (SS): This arm consisted of participants who received stable standard-of-care (SOC) medications at study entry and were randomized to receive dapirolizumab pegol (DZP) 45mg/kg intravenous (iv) infusion every 4 weeks (Q4W) during the 24-week Double-Blind Treatment Period. Participants formed the SS.
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
percentage of participants | 66.7 | 66.7 | 82.2 | 74.5

4. Secondary Outcome: Percentage of Participants With a Serious Adverse Event (SAE)
Description: A Serious Adverse Event (SAE) must have met 1 or more of the following criteria:
  * Death
  * Life threatening
  * Significant or persistent disability/incapacity
  * Congenital anomaly/birth defect (including that occurring in a fetus)
  * Important medical event that, based upon appropriate medical judgment, may have jeopardized the study participant, and may have required medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious
  * Initial inpatient hospitalization or prolongation of hospitalization.
Time Frame: From Baseline (Week 1) until end of the study (Week 48)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
percentage of participants | 13.3 | 11.1 | 13.3 | 10.6

5. Secondary Outcome: Percentage of Participants With at Least One Adverse Events (AEs) of Interest
Description: Adverse events of interest (AEOI) were identified by the Investigator based on definitions per protocol, documented on the electronic Case Report Form (eCRF), adequately monitored, and source controlled.
  AEOI (regardless of seriousness):
  * Moderate to severe infections, including opportunistic infections and tuberculosis (TB)
  * Infusion reactions (including hypersensitivity and anaphylaxis)
  * Thromboembolic events (including but not limited to cardiovascular events, stroke, myocardial infarction, pulmonary embolism, and deep vein thrombosis)
  * Prespecified neurological events: severe and/or serious headache, positional headache, cranial nerve dysfunction, or signs and symptoms of meningitis (photophobia, neck stiffness)
  * Malignancies.
Time Frame: From Baseline (Week 1) until end of the study (Week 48)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
percentage of participants | 24.4 | 26.7 | 28.9 | 25.5

6. Secondary Outcome: Percentage of Participants Who Permanently Withdrew of Study Drug Due to an Adverse Event (AE)
Description: as for outcome 3
Time Frame: From Baseline (Week 1) until end of the study (Week 48)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
percentage of participants | 8.9 | 0 | 4.4 | 4.3

7. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure
Description: Blood pressure was measured in millimetre of mercury (mmHg).
Time Frame: From Baseline (Week 1) to Week 48
Population: The Safety Set (SS) consisted of all study participants who were randomized and received at least 1 dose (any amount) of study drug. Here, 'n' (Number analyzed) signifies participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmHg
  Week 2: number analyzed (Participants) | 45 | 45 | 45 | 44
  Week 2 | 3.3 (12.9) | 5.1 (10.5) | 0.7 (10.7) | 3.2 (9.9)
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | 0.6 (10.8) | 1.0 (7.9) | -2.0 (8.9) | 0.6 (12.4)
  Week 6: number analyzed (Participants) | 43 | 45 | 44 | 45
  Week 6 | 0.3 (11.5) | 4.0 (9.9) | 2.3 (11.0) | 2.4 (10.6)
  Week 8: number analyzed (Participants) | 44 | 44 | 44 | 43
  Week 8 | 0.5 (12.4) | 3.3 (12.6) | -2.4 (9.9) | -0.7 (11.9)
  Week 12: number analyzed (Participants) | 44 | 45 | 45 | 44
  Week 12 | -0.7 (10.1) | 3.2 (10.5) | -3.0 (11.8) | 0.8 (9.2)
  Week 16: number analyzed (Participants) | 43 | 44 | 43 | 44
  Week 16 | 2.1 (12.3) | 2.1 (11.6) | -2.8 (10.6) | 0.9 (11.1)
  Week 20: number analyzed (Participants) | 42 | 45 | 42 | 44
  Week 20 | 1.6 (9.9) | 2.6 (9.8) | -1.7 (12.3) | 1.5 (11.3)
  Week 24: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 24 | -0.7 (14.3) | 1.1 (13.1) | 0.3 (11.0) | 3.6 (9.3)
  Week 28: number analyzed (Participants) | 44 | 43 | 42 | 44
  Week 28 | 1.8 (12.3) | 3.7 (13.1) | 0.9 (10.5) | 2.5 (11.8)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 2.2 (11.1) | 3.0 (13.2) | 0.4 (11.3) | 4.3 (13.7)
  Week 36: number analyzed (Participants) | 42 | 42 | 41 | 41
  Week 36 | 2.1 (11.0) | 3.1 (12.6) | 0.2 (10.5) | 2.4 (12.9)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -1.0 (14.1) | 6.2 (12.9) | -2.0 (11.7) | 2.5 (11.3)
  Week 44: number analyzed (Participants) | 39 | 41 | 41 | 42
  Week 44 | 0.1 (12.6) | 3.3 (14.1) | 1.3 (10.4) | 4.2 (11.8)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 42
  Week 48 | -1.5 (11.5) | 4.9 (14.3) | 0.1 (10.2) | 4.4 (12.0)

8. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure
Description: Blood pressure was measured in millimetre of mercury (mmHg).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmHg
  Week 2: number analyzed (Participants) | 45 | 45 | 45 | 44
  Week 2 | 2.1 (10.5) | 1.4 (8.6) | 1.5 (9.3) | 2.4 (8.2)
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | -0.7 (7.8) | -1.5 (6.3) | -1.7 (8.2) | -0.1 (8.3)
  Week 6: number analyzed (Participants) | 43 | 45 | 44 | 45
  Week 6 | 1.0 (10.0) | 1.5 (8.6) | 1.8 (10.0) | 1.9 (7.9)
  Week 8: number analyzed (Participants) | 44 | 44 | 44 | 43
  Week 8 | 1.1 (9.2) | 0.4 (9.1) | 0.1 (8.6) | 1.0 (8.0)
  Week 12: number analyzed (Participants) | 44 | 45 | 45 | 44
  Week 12 | -0.9 (8.4) | -0.3 (6.9) | -2.2 (9.6) | -0.3 (6.9)
  Week 16: number analyzed (Participants) | 43 | 44 | 43 | 44
  Week 16 | -0.3 (8.9) | -1.3 (7.6) | -0.7 (9.5) | -0.1 (7.0)
  Week 20: number analyzed (Participants) | 42 | 45 | 42 | 44
  Week 20 | 1.5 (8.1) | -1.1 (8.7) | -0.7 (9.6) | 0.9 (8.8)
  Week 24: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 24 | 1.9 (11.2) | 1.6 (8.7) | 2.3 (10.7) | 0.6 (8.7)
  Week 28: number analyzed (Participants) | 44 | 43 | 42 | 44
  Week 28 | 1.5 (9.1) | -0.2 (8.8) | 1.4 (8.4) | 2.5 (8.4)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 2.3 (10.1) | 2.8 (9.3) | 0.7 (10.2) | 2.3 (8.1)
  Week 36: number analyzed (Participants) | 42 | 42 | 41 | 41
  Week 36 | 3.4 (9.8) | 1.4 (10.2) | 1.4 (8.4) | 2.2 (8.0)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | 1.0 (9.2) | 2.6 (7.6) | 0.5 (9.9) | 3.6 (8.8)
  Week 44: number analyzed (Participants) | 39 | 41 | 41 | 42
  Week 44 | 0.8 (10.2) | 1.5 (8.1) | 0.4 (9.4) | 2.2 (10.3)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 42
  Week 48 | 1.4 (9.0) | 2.3 (8.8) | 1.1 (9.4) | 2.4 (8.6)

9. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Description: Pulse Rate was measured in beats per minute (beats/min).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
beats/min
  Week 2: number analyzed (Participants) | 45 | 45 | 45 | 44
  Week 2 | -0.2 (8.3) | 0.2 (10.4) | 2.3 (9.7) | -0.9 (10.4)
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | 1.7 (9.6) | 1.5 (8.0) | 0.4 (8.4) | -3.3 (9.7)
  Week 6: number analyzed (Participants) | 43 | 45 | 44 | 45
  Week 6 | -0.7 (10.2) | 0.1 (8.5) | 0.8 (8.9) | -0.6 (8.8)
  Week 8: number analyzed (Participants) | 44 | 44 | 44 | 43
  Week 8 | 1.3 (9.0) | 0.3 (9.2) | 1.4 (10.2) | -2.6 (10.2)
  Week 12: number analyzed (Participants) | 44 | 45 | 45 | 44
  Week 12 | 0.6 (10.3) | 1.1 (9.8) | -0.3 (10.4) | -1.5 (9.7)
  Week 16: number analyzed (Participants) | 43 | 44 | 43 | 44
  Week 16 | -0.8 (9.2) | 0.3 (8.9) | 0.9 (10.7) | -1.6 (10.6)
  Week 20: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 20 | 0.3 (10.6) | 1.1 (9.9) | 0.8 (9.5) | 0.4 (6.6)
  Week 24: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 24 | -1.5 (10.7) | 0.8 (10.9) | -0.3 (10.2) | -1.0 (8.7)
  Week 28: number analyzed (Participants) | 44 | 43 | 42 | 44
  Week 28 | 0.6 (11.8) | 1.3 (10.9) | 0.0 (9.2) | 0.6 (8.8)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 0.4 (9.8) | 1.3 (10.9) | 0.8 (11.4) | -2.1 (11.0)
  Week 36: number analyzed (Participants) | 42 | 42 | 41 | 41
  Week 36 | -0.7 (10.9) | 0.2 (8.3) | 0.7 (10.4) | -0.2 (9.8)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -0.1 (10.9) | -0.1 (9.8) | 0.6 (10.2) | -1.3 (9.6)
  Week 44: number analyzed (Participants) | 39 | 41 | 41 | 42
  Week 44 | -0.2 (10.2) | -0.1 (9.8) | 0.3 (11.7) | -0.6 (8.9)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 42
  Week 48 | -0.2 (11.1) | -0.7 (10.6) | -0.9 (11.9) | -2.0 (7.7)

10. Secondary Outcome: Mean Change From Baseline in Temperature
Description: Temperature was measured in Grad Celsius (°C).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Temperature (C)
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
Temperature (C)
  Week 2: number analyzed (Participants) | 45 | 45 | 45 | 44
  Week 2 | -0.1 (0.4) | 0.0 (0.3) | 0.1 (0.5) | 0.0 (0.4)
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | -0.1 (0.4) | 0.0 (0.4) | 0.0 (0.4) | 0.0 (0.3)
  Week 6: number analyzed (Participants) | 43 | 45 | 44 | 45
  Week 6 | -0.2 (0.5) | 0.0 (0.4) | 0.1 (0.5) | 0.0 (0.5)
  Week 8: number analyzed (Participants) | 44 | 44 | 44 | 43
  Week 8 | -0.1 (0.4) | -0.1 (0.3) | 0.0 (0.4) | 0.0 (0.4)
  Week 12: number analyzed (Participants) | 44 | 45 | 45 | 44
  Week 12 | -0.1 (0.4) | -0.1 (0.4) | 0.0 (0.3) | 0.0 (0.4)
  Week 16: number analyzed (Participants) | 43 | 44 | 43 | 44
  Week 16 | -0.1 (0.4) | 0.0 (0.4) | 0.0 (0.4) | 0.0 (0.3)
  Week 20: number analyzed (Participants) | 42 | 45 | 42 | 44
  Week 20 | -0.1 (0.4) | 0.0 (0.4) | 0.0 (0.4) | 0.0 (0.5)
  Week 24: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 24 | -0.1 (0.5) | 0.0 (0.4) | 0.1 (0.5) | 0.0 (0.4)
  Week 28: number analyzed (Participants) | 44 | 43 | 42 | 44
  Week 28 | 0.0 (0.4) | 0.0 (0.4) | 0.1 (0.5) | 0.1 (0.5)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 0.0 (0.4) | 0.0 (0.4) | 0.1 (0.5) | 0.0 (0.4)
  Week 36: number analyzed (Participants) | 42 | 42 | 41 | 41
  Week 36 | -0.1 (0.3) | 0.0 (0.6) | 0.0 (0.4) | 0.1 (0.4)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | 0.0 (0.4) | 0.0 (0.4) | 0.0 (0.5) | 0.1 (0.3)
  Week 44: number analyzed (Participants) | 39 | 41 | 41 | 42
  Week 44 | 0.0 (0.6) | 0.0 (0.5) | 0.1 (0.4) | 0.0 (0.4)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 42
  Week 48 | -0.1 (0.4) | 0.0 (0.4) | 0.0 (0.5) | 0.0 (0.4)

11. Secondary Outcome: Mean Change From Baseline in Weight
Description: Weight was measured in kilograms (kg).
Time Frame: Baseline (Week 1), Week 4, Week 8, Week 12, Week 16, and Week 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
kg
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | 0.0 (1.0) | 0.2 (1.0) | 0.4 (0.9) | 0.3 (1.2)
  Week 8: number analyzed (Participants) | 44 | 44 | 43 | 43
  Week 8 | 0.3 (1.9) | 0.6 (1.4) | 0.6 (1.8) | 0.4 (1.8)
  Week 12: number analyzed (Participants) | 43 | 45 | 44 | 44
  Week 12 | 0.4 (2.3) | 0.5 (1.6) | 0.5 (2.0) | 0.6 (2.3)
  Week 16: number analyzed (Participants) | 43 | 44 | 43 | 44
  Week 16 | 0.3 (2.3) | 0.7 (2.3) | 0.8 (2.3) | 0.5 (2.4)
  Week 20: number analyzed (Participants) | 42 | 45 | 42 | 44
  Week 20 | 0.3 (2.4) | 0.7 (2.6) | 1.0 (2.6) | 0.5 (2.8)

12. Secondary Outcome: Mean Change From Baseline in Height
Description: Height was measured in centimeters (cm).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
cm | NA (NA) — Here, 'NA' signifies that height was only measured at Screening as per planned analysis. Therefore, data was not collected for this outcome measure. | NA (NA) — Here, 'NA' signifies that height was only measured at Screening as per planned analysis. Therefore, data was not collected for this outcome measure. | NA (NA) — Here, 'NA' signifies that height was only measured at Screening as per planned analysis. Therefore, data was not collected for this outcome measure. | NA (NA) — Here, 'NA' signifies that height was only measured at Screening as per planned analysis. Therefore, data was not collected for this outcome measure.

13. Secondary Outcome: Number of Participants With 12-Lead Electrocardiogram (ECG) Abnormal Findings
Description: Twelve-lead ECG assessments should have been performed prior to dosing (if applicable) and prior to obtaining pharmacokinetic (PK) or other laboratory samples. Electrocardiograms were recorded digitally and read by the Investigator for recording in the electronic Case Report Form (eCRF).
Time Frame: Screening, Week 4, Week 24, Week 28 and Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
Participants
  Screening | 8 | 11 | 6 | 6
  Week 4 | 11 | 12 | 7 | 10
  Week 24 | 9 | 7 | 6 | 10
  Week 28 | 1 | 0 | 0 | 0
  Week 48 | 8 | 7 | 11 | 9

14. Secondary Outcome: Mean Change From Baseline in Hemoglobin
Description: Hemoglobin was measured in grams per liter (g/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
g/L
  Week 2: number analyzed (Participants) | 44 | 42 | 45 | 42
  Week 2 | 0.4 (6.4) | -1.8 (5.8) | -0.7 (6.9) | -0.7 (6.8)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -1.0 (7.2) | -0.7 (7.7) | -1.4 (8.6) | -0.8 (5.8)
  Week 8: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 8 | -0.3 (7.3) | -1.9 (7.9) | -1.9 (8.6) | -1.3 (7.4)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | -0.5 (9.5) | -0.5 (8.5) | -0.5 (10.1) | 0.2 (8.3)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | 0.3 (10.4) | -0.3 (10.0) | -0.8 (10.6) | -2.7 (8.3)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | -0.7 (11.5) | 0.3 (9.9) | -0.5 (10.1) | -2.4 (7.2)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.4 (9.7) | -0.7 (11.2) | -0.7 (10.5) | -2.9 (8.1)
  Week 28: number analyzed (Participants) | 44 | 41 | 41 | 44
  Week 28 | 0.7 (10.6) | -3.4 (11.0) | 0.0 (14.1) | -3.1 (9.5)
  Week 32: number analyzed (Participants) | 43 | 43 | 43 | 42
  Week 32 | 1.6 (12.5) | -1.3 (9.8) | 1.0 (12.5) | -1.3 (9.6)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | 0.7 (13.5) | -0.3 (13.5) | 1.9 (14.9) | 1.1 (11.0)
  Week 48: number analyzed (Participants) | 38 | 42 | 39 | 42
  Week 48 | -0.5 (14.3) | -1.5 (11.6) | 0.9 (12.5) | -0.7 (10.0)

15. Secondary Outcome: Mean Change From Baseline in Hematocrit
Description: Hematocrit was measured in volume percentage (%) of red blood cells in blood.
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: volume % of red blood cells
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
volume % of red blood cells
  Week 2: number analyzed (Participants) | 44 | 42 | 45 | 42
  Week 2 | 0.42 (2.52) | -0.25 (2.26) | -0.32 (2.37) | 0.00 (2.71)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.46 (2.29) | -0.17 (2.75) | -0.79 (2.92) | -0.11 (2.31)
  Week 8: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 8 | -0.27 (2.23) | -0.12 (2.94) | -0.86 (2.72) | -0.42 (2.31)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | -0.23 (2.67) | -0.13 (2.72) | -0.32 (3.39) | -0.02 (2.54)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | -0.12 (2.86) | 0.05 (3.25) | -0.57 (3.32) | -0.84 (2.95)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | -0.41 (3.20) | 0.13 (2.99) | -0.42 (3.32) | -0.80 (2.83)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.09 (2.61) | -0.40 (3.19) | -0.29 (3.14) | -0.76 (2.33)
  Week 28: number analyzed (Participants) | 44 | 41 | 41 | 44
  Week 28 | 0.03 (2.98) | -1.02 (3.23) | -0.22 (3.99) | -0.89 (2.47)
  Week 32: number analyzed (Participants) | 43 | 43 | 43 | 42
  Week 32 | 0.29 (2.89) | -0.62 (2.86) | 0.17 (3.43) | -0.21 (2.82)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -0.20 (3.32) | -0.24 (4.37) | 0.58 (4.11) | 0.37 (2.72)
  Week 48: number analyzed (Participants) | 38 | 42 | 39 | 42
  Week 48 | -0.59 (3.51) | -0.37 (3.58) | -0.08 (3.21) | -0.11 (2.54)

16. Secondary Outcome: Mean Change From Baseline in Erythrocytes
Description: Erythrocytes was measured in number of erythrocytes per liter (10^12/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^12 erythrocytes per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^12 erythrocytes per liter
  Week 2: number analyzed (Participants) | 44 | 42 | 45 | 42
  Week 2 | -0.004 (0.246) | -0.035 (0.237) | -0.032 (0.223) | -0.028 (0.237)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.080 (0.243) | -0.018 (0.293) | -0.052 (0.273) | -0.033 (0.210)
  Week 8: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 8 | -0.039 (0.224) | -0.039 (0.280) | -0.069 (0.262) | -0.044 (0.242)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | -0.024 (0.271) | 0.014 (0.292) | -0.010 (0.267) | 0.019 (0.226)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | -0.002 (0.312) | 0.041 (0.360) | 0.000 (0.302) | -0.051 (0.265)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | -0.029 (0.333) | 0.062 (0.309) | -0.001 (0.325) | -0.047 (0.302)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 0.005 (0.308) | 0.036 (0.312) | 0.013 (0.319) | -0.038 (0.240)
  Week 28: number analyzed (Participants) | 44 | 41 | 41 | 44
  Week 28 | 0.018 (0.340) | -0.040 (0.304) | 0.019 (0.346) | -0.050 (0.270)
  Week 32: number analyzed (Participants) | 43 | 43 | 43 | 42
  Week 32 | 0.048 (0.320) | 0.001 (0.284) | 0.032 (0.289) | 0.027 (0.277)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -0.005 (0.343) | 0.042 (0.382) | 0.054 (0.368) | 0.060 (0.256)
  Week 48: number analyzed (Participants) | 38 | 42 | 39 | 42
  Week 48 | -0.024 (0.332) | -0.018 (0.295) | 0.017 (0.299) | -0.028 (0.245)

17. Secondary Outcome: Mean Change From Baseline in Erythrocytes Mean Corpuscular Volume
Description: Erythrocytes Mean Corpuscular Volume was measured in femtolitres (fL).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Femtolitres (fL)
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
Femtolitres (fL)
  Week 2: number analyzed (Participants) | 44 | 42 | 45 | 42
  Week 2 | 1.01 (2.28) | 0.24 (2.40) | -0.09 (2.66) | 0.45 (2.96)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.60 (2.35) | 0.08 (2.66) | -0.68 (2.10) | 0.40 (3.02)
  Week 8: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 8 | 0.23 (3.48) | -0.30 (5.36) | -0.54 (2.85) | -0.16 (2.79)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | 0.06 (3.57) | -0.52 (3.44) | -0.55 (4.67) | -0.57 (3.09)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | -0.25 (3.41) | -0.65 (4.38) | -1.38 (4.87) | -0.97 (3.62)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | -0.37 (3.73) | -0.92 (4.58) | -1.00 (5.01) | -0.97 (3.54)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.23 (3.83) | -1.63 (4.07) | -0.92 (6.51) | -1.05 (4.00)
  Week 28: number analyzed (Participants) | 44 | 41 | 41 | 44
  Week 28 | -0.33 (3.61) | -1.40 (4.61) | -0.96 (6.46) | -1.21 (4.91)
  Week 32: number analyzed (Participants) | 43 | 43 | 43 | 42
  Week 32 | -0.27 (4.45) | -1.33 (4.32) | -0.45 (6.81) | -1.06 (4.69)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -0.36 (5.34) | -1.46 (4.72) | 0.07 (6.27) | -0.24 (4.85)
  Week 48: number analyzed (Participants) | 38 | 42 | 39 | 42
  Week 48 | -0.98 (5.34) | -0.50 (4.97) | -0.63 (6.92) | 0.34 (4.31)

18. Secondary Outcome: Mean Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration
Description: Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration was measured in grams per liter (g/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
g/L
  Week 2: number analyzed (Participants) | 44 | 42 | 45 | 42
  Week 2 | -2.3 (9.8) | -2.6 (10.9) | 0.7 (9.8) | -1.9 (10.1)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 1.4 (8.7) | -0.9 (10.1) | 2.7 (8.6) | -1.2 (12.5)
  Week 8: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 8 | 1.7 (11.5) | -3.8 (13.4) | 2.1 (8.2) | -0.1 (11.5)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | 0.5 (11.1) | -0.6 (10.7) | 0.6 (12.3) | 0.5 (12.7)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | 1.6 (13.8) | -1.5 (10.1) | 2.3 (11.3) | -0.2 (14.1)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | 1.6 (12.9) | -0.9 (11.3) | 2.4 (11.2) | 0.4 (12.6)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 0.0 (13.7) | 1.0 (13.2) | 0.4 (12.8) | -1.2 (13.1)
  Week 28: number analyzed (Participants) | 44 | 41 | 41 | 44
  Week 28 | 1.6 (13.4) | -1.3 (14.4) | 1.7 (13.8) | -0.6 (16.5)
  Week 32: number analyzed (Participants) | 43 | 43 | 43 | 42
  Week 32 | 1.7 (18.9) | 1.1 (13.8) | 1.2 (15.0) | -1.4 (16.0)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | 3.4 (17.6) | 0.8 (16.5) | 0.1 (15.8) | 0.1 (15.4)
  Week 48: number analyzed (Participants) | 38 | 42 | 39 | 42
  Week 48 | 3.6 (17.1) | -0.6 (16.2) | 2.9 (14.5) | 0.0 (13.5)

19. Secondary Outcome: Mean Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin
Description: Erythrocytes Mean Corpuscular Hemoglobin was measured in picograms (pg).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
Picograms (pg)
  Week 2: number analyzed (Participants) | 44 | 42 | 45 | 42
  Week 2 | 0.12 (0.71) | -0.18 (0.65) | 0.04 (0.43) | 0.00 (0.47)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.31 (0.63) | -0.06 (0.79) | 0.04 (0.64) | 0.02 (0.65)
  Week 8: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 8 | 0.20 (0.87) | -0.25 (0.87) | 0.04 (0.81) | -0.04 (0.74)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | 0.04 (1.08) | -0.25 (1.03) | -0.09 (1.25) | -0.12 (0.90)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | 0.03 (1.43) | -0.36 (1.31) | -0.20 (1.52) | -0.31 (1.19)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | 0.00 (1.49) | -0.39 (1.40) | -0.10 (1.63) | -0.26 (1.24)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.13 (1.57) | -0.43 (1.39) | -0.25 (1.96) | -0.44 (1.42)
  Week 28: number analyzed (Participants) | 44 | 41 | 41 | 44
  Week 28 | 0.01 (1.68) | -0.55 (1.45) | -0.15 (2.09) | -0.44 (1.68)
  Week 32: number analyzed (Participants) | 43 | 43 | 43 | 42
  Week 32 | 0.01 (2.12) | -0.33 (1.28) | -0.06 (2.39) | -0.48 (1.63)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | 0.17 (2.50) | -0.40 (1.30) | 0.03 (2.32) | -0.09 (2.00)
  Week 48: number analyzed (Participants) | 38 | 42 | 39 | 42
  Week 48 | 0.02 (2.58) | -0.21 (1.48) | 0.06 (2.55) | 0.10 (1.90)

20. Secondary Outcome: Mean Change From Baseline in Leukocytes
Description: Leukocytes was measured in number of leukocytes per liter (10^9/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 leukocytes per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^9 leukocytes per liter
  Week 2: number analyzed (Participants) | 44 | 42 | 45 | 42
  Week 2 | 0.34 (2.45) | 0.27 (1.23) | 0.49 (1.46) | 0.20 (1.62)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.10 (1.88) | 0.27 (1.63) | 0.25 (1.47) | 0.52 (2.11)
  Week 8: number analyzed (Participants) | 43 | 44 | 44 | 44
  Week 8 | -0.25 (2.12) | 0.46 (1.41) | -0.05 (1.50) | -0.10 (1.65)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 43
  Week 12 | -0.27 (1.80) | 0.18 (1.73) | 0.17 (2.00) | 0.23 (2.01)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | -0.31 (2.18) | 0.13 (1.55) | 0.21 (1.69) | -0.20 (2.12)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | -0.24 (2.27) | -0.06 (1.59) | -0.22 (1.74) | 0.30 (2.61)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.22 (2.41) | -0.12 (1.83) | -0.14 (1.75) | -0.34 (1.97)
  Week 28: number analyzed (Participants) | 44 | 41 | 41 | 44
  Week 28 | 0.05 (2.04) | 0.06 (1.93) | 0.26 (2.04) | -0.58 (1.70)
  Week 32: number analyzed (Participants) | 43 | 43 | 43 | 42
  Week 32 | -0.14 (2.20) | 0.08 (1.64) | 0.19 (1.67) | -0.44 (1.68)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | 0.17 (2.54) | 0.04 (1.60) | -0.35 (1.49) | -0.49 (1.96)
  Week 48: number analyzed (Participants) | 38 | 42 | 39 | 42
  Week 48 | -0.49 (1.83) | 0.30 (1.53) | -0.14 (2.06) | -0.62 (1.87)

21. Secondary Outcome: Mean Change From Baseline in Basophils
Description: Basophils was measured in number of basophils per liter (10^9/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 basophils per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^9 basophils per liter
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | 0.01 (0.03) | 0.02 (0.04) | 0.00 (0.03) | 0.00 (0.02)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | 0.01 (0.03) | 0.00 (0.03) | 0.01 (0.04) | 0.00 (0.02)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | 0.01 (0.04) | 0.01 (0.04) | 0.01 (0.03) | 0.00 (0.02)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | 0.01 (0.03) | 0.01 (0.04) | 0.00 (0.03) | 0.00 (0.03)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | 0.01 (0.04) | 0.00 (0.03) | 0.01 (0.03) | 0.00 (0.03)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | 0.00 (0.03) | 0.01 (0.03) | 0.00 (0.03) | 0.00 (0.03)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | 0.00 (0.03) | 0.02 (0.04) | 0.00 (0.03) | 0.00 (0.03)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | 0.02 (0.05) | 0.01 (0.04) | 0.00 (0.02) | 0.00 (0.03)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | 0.00 (0.03) | 0.00 (0.02) | 0.01 (0.03) | 0.00 (0.03)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | 0.00 (0.02) | 0.00 (0.02) | 0.01 (0.03) | 0.00 (0.03)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | 0.00 (0.03) | 0.00 (0.02) | 0.00 (0.03) | 0.01 (0.03)

22. Secondary Outcome: Mean Change From Baseline in Basophils/Leukocytes
Description: Basophils/Leukocytes was measured in percentages (%).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of Basophils per Leukocytes
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of Basophils per Leukocytes
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | -0.05 (0.23) | 0.02 (0.20) | -0.05 (0.31) | -0.03 (0.27)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | 0.03 (0.27) | -0.06 (0.26) | -0.01 (0.43) | -0.07 (0.26)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | 0.08 (0.42) | 0.03 (0.32) | 0.00 (0.33) | -0.06 (0.23)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | 0.04 (0.30) | 0.09 (0.48) | 0.00 (0.25) | -0.07 (0.28)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | 0.01 (0.25) | 0.00 (0.28) | -0.02 (0.31) | -0.05 (0.30)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | -0.02 (0.26) | 0.00 (0.27) | -0.07 (0.29) | -0.04 (0.32)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | -0.04 (0.31) | 0.15 (0.44) | -0.03 (0.24) | -0.03 (0.21)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | 0.08 (0.54) | 0.03 (0.29) | 0.00 (0.24) | 0.07 (0.32)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | -0.03 (0.29) | 0.00 (0.23) | 0.01 (0.25) | 0.01 (0.25)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | -0.08 (0.24) | -0.03 (0.25) | 0.07 (0.29) | 0.01 (0.29)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | -0.01 (0.29) | -0.08 (0.21) | 0.02 (0.25) | 0.06 (0.28)

23. Secondary Outcome: Mean Change From Baseline in Eosinophils
Description: Eosinophils was measured in number of eosinophils per liter (10^9/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 eosinophils per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^9 eosinophils per liter
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | -0.01 (0.04) | 0.01 (0.06) | 0.00 (0.09) | -0.01 (0.05)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | -0.01 (0.04) | -0.01 (0.06) | 0.00 (0.04) | -0.01 (0.04)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | -0.01 (0.04) | 0.03 (0.16) | 0.00 (0.04) | 0.01 (0.07)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | 0.00 (0.04) | 0.04 (0.20) | 0.02 (0.10) | 0.02 (0.17)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | 0.00 (0.05) | 0.02 (0.11) | 0.01 (0.05) | 0.00 (0.06)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | 0.00 (0.05) | 0.04 (0.24) | 0.01 (0.05) | -0.01 (0.05)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | -0.01 (0.05) | 0.04 (0.15) | 0.02 (0.07) | -0.02 (0.06)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | -0.01 (0.04) | 0.01 (0.07) | 0.01 (0.05) | 0.00 (0.06)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | -0.01 (0.06) | 0.01 (0.10) | 0.01 (0.05) | -0.02 (0.04)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | 0.00 (0.05) | 0.01 (0.06) | 0.02 (0.06) | 0.00 (0.07)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | 0.00 (0.04) | -0.01 (0.05) | 0.00 (0.06) | 0.00 (0.06)

24. Secondary Outcome: Mean Change From Baseline in Eosinophils/Leukocytes
Description: Eosinophils/Leukocytes was measured in percentages (%).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of Eosinophils per Leukocytes
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of Eosinophils per Leukocytes
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | -0.19 (1.07) | 0.07 (0.86) | -0.18 (1.13) | -0.29 (1.22)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | -0.32 (0.96) | -0.05 (1.26) | -0.12 (1.01) | -0.26 (0.94)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | -0.05 (1.09) | 0.54 (2.13) | 0.10 (1.11) | 0.22 (1.89)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | 0.18 (1.03) | 0.70 (3.12) | 0.33 (1.68) | 0.05 (1.83)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | 0.06 (1.05) | 0.36 (1.24) | 0.20 (1.40) | -0.11 (1.33)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | 0.04 (1.11) | 0.83 (3.58) | 0.11 (1.24) | -0.39 (1.29)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | 0.11 (1.16) | 0.82 (2.89) | -0.01 (1.22) | 0.06 (1.63)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | 0.06 (1.00) | 0.21 (1.33) | 0.18 (1.02) | -0.03 (1.35)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | 0.02 (1.09) | 0.28 (1.60) | 0.16 (1.13) | -0.20 (1.03)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | -0.10 (0.85) | 0.05 (1.09) | 0.40 (1.23) | -0.09 (1.47)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | 0.09 (1.02) | -0.17 (1.08) | 0.06 (0.90) | 0.24 (1.03)

25. Secondary Outcome: Mean Change From Baseline in Lymphocytes
Description: Lymphocytes was measured in number of lymphocytes per liter (10^9/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 lymphocytes per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^9 lymphocytes per liter
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | -0.03 (0.39) | 0.05 (0.36) | 0.16 (0.29) | 0.24 (0.37)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | -0.04 (0.36) | -0.01 (0.47) | -0.01 (0.41) | 0.23 (0.42)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | -0.15 (0.48) | -0.03 (0.39) | 0.06 (0.46) | 0.14 (0.50)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | -0.06 (0.43) | 0.02 (0.59) | 0.01 (0.42) | 0.21 (0.51)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | -0.09 (0.52) | -0.11 (0.51) | -0.02 (0.47) | 0.04 (0.40)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | -0.14 (0.56) | -0.13 (0.54) | 0.02 (0.39) | 0.13 (0.55)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | -0.11 (0.51) | -0.08 (0.60) | -0.03 (0.45) | 0.05 (0.52)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | -0.04 (0.57) | -0.02 (0.59) | 0.01 (0.53) | 0.03 (0.56)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | -0.11 (0.57) | -0.16 (0.59) | 0.05 (0.45) | -0.02 (0.44)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | -0.11 (0.54) | -0.11 (0.52) | -0.11 (0.43) | -0.03 (0.48)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | -0.19 (0.68) | -0.19 (0.60) | -0.10 (0.44) | -0.02 (0.49)

26. Secondary Outcome: Mean Change From Baseline in Lymphocytes/Leukocytes
Description: Lymphocytes/Leukocytes was measured in percentages (%).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of Lymphocytes per Leukocytes
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of Lymphocytes per Leukocytes
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | -1.88 (9.01) | 0.19 (6.55) | 1.18 (6.09) | 2.61 (6.11)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | -0.88 (7.09) | -1.02 (6.34) | -1.18 (9.93) | 0.97 (8.00)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | -1.98 (10.59) | -1.40 (7.13) | 0.56 (10.20) | 1.97 (8.51)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | 0.21 (7.87) | 0.56 (10.58) | -0.44 (9.90) | 2.46 (10.18)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | -0.91 (8.33) | -1.49 (7.50) | -1.18 (9.65) | 0.12 (9.34)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | -1.97 (10.37) | -0.66 (6.58) | 0.88 (10.69) | 0.71 (10.32)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | -0.75 (8.69) | -0.56 (7.35) | -0.52 (10.55) | 1.85 (9.67)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | -1.18 (8.27) | -0.05 (8.51) | -0.05 (9.97) | 1.61 (10.55)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | -1.59 (7.69) | -2.56 (6.51) | -0.16 (7.70) | 0.70 (8.74)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | -2.60 (9.18) | -2.02 (5.99) | -1.36 (10.12) | 0.33 (8.41)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | -1.46 (11.29) | -3.71 (7.41) | -0.84 (9.42) | 1.69 (10.05)

27. Secondary Outcome: Mean Change From Baseline in Monocytes
Description: Monocytes was measured in number of monocytes per liter (10^9/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 monocytes per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^9 monocytes per liter
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | -0.01 (0.17) | 0.01 (0.18) | 0.05 (0.14) | 0.01 (0.13)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | 0.01 (0.18) | 0.04 (0.18) | 0.01 (0.14) | 0.06 (0.19)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | -0.03 (0.18) | 0.04 (0.18) | 0.03 (0.16) | 0.02 (0.17)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | -0.01 (0.19) | 0.00 (0.14) | 0.04 (0.18) | 0.06 (0.15)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | -0.01 (0.17) | 0.01 (0.17) | 0.05 (0.18) | 0.03 (0.14)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | -0.03 (0.19) | 0.00 (0.16) | 0.00 (0.13) | 0.05 (0.19)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | 0.00 (0.19) | 0.04 (0.19) | 0.03 (0.17) | 0.00 (0.17)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | 0.00 (0.20) | 0.04 (0.21) | 0.08 (0.19) | 0.02 (0.17)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | -0.01 (0.18) | 0.02 (0.19) | 0.05 (0.23) | -0.01 (0.19)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | 0.03 (0.17) | 0.05 (0.16) | 0.04 (0.16) | -0.01 (0.18)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | -0.02 (0.20) | -0.01 (0.13) | 0.03 (0.15) | -0.02 (0.18)

28. Secondary Outcome: Mean Change From Baseline in Monocytes/Leukocytes
Description: Monocytes/Leukocytes was measured in percentages (%).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of Monocytes per Leukocytes
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of Monocytes per Leukocytes
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | -0.87 (2.50) | -0.07 (2.46) | 0.23 (3.03) | -0.37 (2.25)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | 0.26 (3.30) | 0.27 (2.41) | -0.16 (3.11) | -0.24 (2.82)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | -0.21 (3.47) | 0.07 (3.61) | 0.51 (3.83) | 0.08 (3.12)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | 0.07 (2.79) | -0.11 (2.38) | 0.22 (3.37) | 0.45 (2.74)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | 0.06 (3.30) | 0.59 (2.85) | 0.43 (3.31) | 0.28 (3.13)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | -0.27 (3.84) | 0.56 (3.08) | 0.33 (3.81) | 0.43 (3.39)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | 0.06 (3.45) | 0.84 (2.97) | 0.46 (3.00) | 0.41 (3.24)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | -0.24 (3.54) | 0.69 (3.24) | 0.64 (3.67) | 0.94 (3.78)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | -0.08 (3.11) | 0.13 (2.62) | 0.46 (3.91) | -0.03 (3.76)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | 0.49 (3.55) | 0.64 (2.92) | 0.83 (3.69) | 0.59 (3.07)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | -0.04 (3.79) | -0.13 (2.41) | 0.47 (3.82) | 0.29 (3.30)

29. Secondary Outcome: Mean Change From Baseline in Neutrophils
Description: Neutrophils was measured in number of neutrophils per liter (10^9/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 neutrophils per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^9 neutrophils per liter
  Week 2: number analyzed (Participants) | 43 | 39 | 44 | 41
  Week 2 | 0.28 (2.43) | 0.26 (1.17) | 0.17 (1.33) | -0.01 (1.46)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | 0.07 (1.82) | 0.27 (1.40) | 0.21 (1.64) | 0.23 (1.96)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | -0.13 (2.20) | 0.41 (1.32) | -0.07 (1.53) | -0.20 (1.49)
  Week 12: number analyzed (Participants) | 44 | 41 | 44 | 42
  Week 12 | -0.24 (1.56) | 0.20 (1.65) | 0.10 (1.94) | -0.01 (2.03)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | -0.22 (2.13) | 0.20 (1.41) | 0.15 (1.61) | -0.20 (2.14)
  Week 20: number analyzed (Participants) | 42 | 41 | 40 | 42
  Week 20 | -0.07 (2.21) | 0.01 (1.22) | -0.39 (1.69) | 0.09 (2.51)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | -0.12 (2.24) | -0.06 (1.54) | -0.16 (1.77) | -0.38 (1.92)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | 0.04 (1.81) | 0.13 (1.64) | 0.10 (1.91) | -0.62 (1.78)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | -0.07 (1.87) | 0.33 (1.27) | 0.07 (1.54) | -0.40 (1.67)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | 0.16 (2.37) | 0.16 (1.31) | -0.32 (1.57) | -0.41 (1.88)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | -0.29 (1.58) | 0.55 (1.15) | -0.09 (2.02) | -0.54 (1.78)

30. Secondary Outcome: Mean Change From Baseline in Neutrophils/Leukocytes
Description: Neutrophils/Leukocytes was measured in percentages (%).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of Neutrophils per Leukocytes
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of Neutrophils per Leukocytes
  Week 2: number analyzed (Participants) | 42 | 39 | 44 | 41
  Week 2 | 2.99 (10.73) | -0.21 (7.94) | -1.20 (8.40) | -1.93 (8.18)
  Week 4: number analyzed (Participants) | 43 | 43 | 41 | 46
  Week 4 | 0.91 (9.37) | 0.89 (7.82) | 1.47 (12.70) | -0.37 (10.27)
  Week 8: number analyzed (Participants) | 42 | 41 | 43 | 43
  Week 8 | 2.15 (12.95) | 0.79 (8.80) | -1.17 (13.28) | -2.23 (10.92)
  Week 12: number analyzed (Participants) | 44 | 40 | 44 | 42
  Week 12 | -0.52 (9.44) | -1.25 (11.78) | -0.12 (13.18) | -2.90 (12.85)
  Week 16: number analyzed (Participants) | 43 | 42 | 43 | 44
  Week 16 | 0.77 (11.02) | 0.54 (8.50) | 0.56 (12.48) | -0.24 (12.23)
  Week 20: number analyzed (Participants) | 42 | 40 | 40 | 42
  Week 20 | 2.22 (13.21) | -0.73 (8.42) | -1.25 (14.29) | -0.71 (13.91)
  Week 24: number analyzed (Participants) | 41 | 40 | 44 | 44
  Week 24 | 0.65 (11.48) | -1.25 (8.74) | 0.10 (13.20) | -2.30 (12.41)
  Week 28: number analyzed (Participants) | 44 | 39 | 40 | 44
  Week 28 | 1.28 (10.38) | -0.88 (10.56) | -0.77 (13.27) | -2.60 (13.79)
  Week 32: number analyzed (Participants) | 41 | 40 | 43 | 42
  Week 32 | 1.67 (9.93) | 2.15 (7.42) | -0.47 (9.80) | -0.48 (12.08)
  Week 40: number analyzed (Participants) | 41 | 42 | 40 | 43
  Week 40 | 2.29 (11.66) | 1.36 (6.95) | 0.07 (13.23) | -0.93 (11.50)
  Week 48: number analyzed (Participants) | 37 | 41 | 39 | 41
  Week 48 | 1.41 (13.58) | 4.09 (8.40) | 0.30 (12.47) | -2.28 (12.38)

31. Secondary Outcome: Mean Change From Baseline in Platelets
Description: Platelets was measured in number of platelets per liter (10^9/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
10^9 platelets per liter
  Week 2: number analyzed (Participants) | 41 | 42 | 45 | 42
  Week 2 | 5.9 (33.2) | 10.0 (40.0) | 1.4 (47.5) | -1.0 (52.0)
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | -5.2 (51.3) | 0.0 (32.4) | 4.9 (43.8) | 8.1 (42.6)
  Week 8: number analyzed (Participants) | 42 | 44 | 44 | 44
  Week 8 | 0.2 (45.3) | -0.3 (40.3) | 3.9 (52.0) | -6.4 (40.5)
  Week 12: number analyzed (Participants) | 43 | 43 | 43 | 44
  Week 12 | -4.3 (50.6) | -1.7 (38.8) | -2.7 (49.0) | 1.8 (49.4)
  Week 16: number analyzed (Participants) | 44 | 43 | 43 | 45
  Week 16 | 0.7 (57.7) | -0.7 (40.5) | -1.5 (66.7) | -2.3 (68.1)
  Week 20: number analyzed (Participants) | 42 | 43 | 41 | 42
  Week 20 | 9.2 (57.1) | -3.3 (43.0) | 0.5 (44.6) | 0.8 (64.4)
  Week 24: number analyzed (Participants) | 42 | 41 | 44 | 43
  Week 24 | 0.2 (60.2) | -5.2 (43.8) | 2.4 (68.6) | 1.7 (67.0)
  Week 28: number analyzed (Participants) | 42 | 41 | 41 | 44
  Week 28 | 3.6 (64.6) | 1.8 (52.6) | -5.8 (71.9) | 1.5 (64.4)
  Week 32: number analyzed (Participants) | 42 | 42 | 42 | 40
  Week 32 | 4.0 (71.8) | -1.9 (55.4) | -4.6 (57.5) | 9.9 (93.8)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 43
  Week 40 | 10.3 (74.9) | 14.2 (52.7) | -8.8 (63.2) | -1.5 (67.4)
  Week 48: number analyzed (Participants) | 37 | 42 | 39 | 42
  Week 48 | 7.1 (67.4) | 3.5 (58.2) | -9.5 (70.9) | -8.8 (66.5)

32. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation 3 (CD3)
Description: Cluster of differentiation 3 (CD3) was measured in cells per microliter (cells/µL).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
cells/µL
  Week 2: number analyzed (Participants) | 38 | 40 | 42 | 40
  Week 2 | 33.0 (313.6) | 77.7 (383.6) | 106.6 (283.1) | 126.9 (338.9)
  Week 4: number analyzed (Participants) | 39 | 40 | 40 | 39
  Week 4 | -30.6 (293.5) | -47.7 (504.3) | 24.0 (394.9) | 227.2 (412.1)
  Week 8: number analyzed (Participants) | 38 | 40 | 39 | 40
  Week 8 | -64.7 (405.7) | -58.6 (422.8) | -20.5 (403.2) | 78.3 (560.0)
  Week 12: number analyzed (Participants) | 41 | 41 | 40 | 40
  Week 12 | -44.2 (283.2) | -48.8 (452.1) | -57.8 (385.1) | 43.7 (599.3)
  Week 16: number analyzed (Participants) | 38 | 42 | 38 | 42
  Week 16 | -81.9 (479.4) | -141.2 (516.1) | -4.5 (383.2) | -45.4 (520.8)
  Week 20: number analyzed (Participants) | 40 | 40 | 39 | 42
  Week 20 | -92.7 (391.1) | -173.4 (490.9) | 5.9 (352.9) | -89.9 (577.7)
  Week 24: number analyzed (Participants) | 39 | 39 | 42 | 43
  Week 24 | -85.8 (472.5) | -128.9 (569.4) | -88.5 (462.1) | -78.3 (570.7)
  Week 28: number analyzed (Participants) | 41 | 40 | 39 | 38
  Week 28 | -27.6 (507.3) | -81.2 (652.7) | 46.1 (482.2) | 7.4 (561.2)
  Week 32: number analyzed (Participants) | 41 | 41 | 41 | 41
  Week 32 | -70.9 (428.4) | -173.6 (565.8) | 18.0 (415.0) | -90.5 (504.0)
  Week 40: number analyzed (Participants) | 40 | 41 | 39 | 43
  Week 40 | -110.5 (526.4) | -166.9 (542.2) | -1.8 (410.7) | 31.7 (528.8)
  Week 48: number analyzed (Participants) | 35 | 40 | 35 | 41
  Week 48 | -115.6 (581.1) | -253.1 (637.0) | 36.1 (492.3) | 22.3 (558.0)

33. Secondary Outcome: Mean Change From Baseline in CD3/Lymphocytes
Description: CD3/Lymphocytes was measured in percentages (%).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of CD3 per Leukocytes
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of CD3 per Leukocytes
  Week 2: number analyzed (Participants) | 38 | 40 | 42 | 40
  Week 2 | -0.7 (6.1) | -0.9 (4.6) | -2.0 (5.7) | -0.2 (7.8)
  Week 4: number analyzed (Participants) | 39 | 40 | 40 | 39
  Week 4 | -2.1 (7.3) | -0.5 (6.0) | -1.9 (5.0) | -0.5 (6.8)
  Week 8: number analyzed (Participants) | 38 | 40 | 39 | 40
  Week 8 | -0.9 (6.1) | -1.2 (4.8) | -2.6 (5.9) | 0.6 (9.5)
  Week 12: number analyzed (Participants) | 41 | 41 | 40 | 40
  Week 12 | -0.4 (5.6) | -1.1 (8.2) | -2.4 (6.0) | -0.1 (9.2)
  Week 16: number analyzed (Participants) | 38 | 42 | 38 | 42
  Week 16 | -1.9 (5.8) | -1.6 (7.8) | -1.9 (7.6) | -1.4 (7.9)
  Week 20: number analyzed (Participants) | 40 | 40 | 39 | 42
  Week 20 | -0.8 (5.0) | 0.0 (8.6) | -2.3 (6.9) | 0.6 (9.2)
  Week 24: number analyzed (Participants) | 39 | 39 | 42 | 43
  Week 24 | 0.0 (6.5) | -0.1 (8.8) | -1.8 (6.6) | 18.7 (114.3)
  Week 28: number analyzed (Participants) | 41 | 40 | 39 | 38
  Week 28 | -0.2 (6.9) | 0.2 (8.3) | -2.9 (7.2) | 0.9 (10.2)
  Week 32: number analyzed (Participants) | 41 | 41 | 41 | 41
  Week 32 | -1.3 (7.0) | 0.2 (7.9) | -1.8 (6.8) | 1.4 (8.5)
  Week 40: number analyzed (Participants) | 40 | 41 | 39 | 43
  Week 40 | 0.2 (6.7) | 1.4 (6.9) | 0.5 (6.5) | 3.3 (7.9)
  Week 48: number analyzed (Participants) | 35 | 40 | 35 | 41
  Week 48 | 1.3 (8.0) | 0.3 (7.6) | 0.1 (6.2) | 4.5 (7.3)

34. Secondary Outcome: Mean Change From Baseline in Cluster of Differentiation 19 (CD19)
Description: Cluster of differentiation 19 (CD19) was measured in cells per microliter (cells/µL).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
cells/µL
  Week 2: number analyzed (Participants) | 38 | 40 | 42 | 40
  Week 2 | 9.6 (56.7) | 12.3 (76.2) | 24.8 (71.0) | 63.4 (133.5)
  Week 4: number analyzed (Participants) | 39 | 40 | 40 | 39
  Week 4 | -2.8 (46.3) | -31.2 (177.0) | 9.2 (60.5) | 82.8 (154.5)
  Week 8: number analyzed (Participants) | 38 | 40 | 39 | 40
  Week 8 | -13.3 (72.9) | -29.4 (183.5) | 8.7 (70.8) | 19.4 (146.4)
  Week 12: number analyzed (Participants) | 41 | 41 | 40 | 40
  Week 12 | -2.6 (83.4) | -48.1 (207.1) | -17.9 (77.8) | 53.2 (203.6)
  Week 16: number analyzed (Participants) | 38 | 42 | 38 | 42
  Week 16 | -12.5 (84.3) | -50.1 (201.5) | -10.0 (92.4) | 13.2 (147.8)
  Week 20: number analyzed (Participants) | 40 | 40 | 39 | 42
  Week 20 | -15.1 (86.0) | -75.4 (216.6) | -2.5 (57.1) | 2.7 (132.6)
  Week 24: number analyzed (Participants) | 39 | 39 | 42 | 43
  Week 24 | -15.0 (89.3) | -77.2 (231.9) | -20.3 (72.0) | -1.1 (135.0)
  Week 28: number analyzed (Participants) | 41 | 40 | 39 | 38
  Week 28 | -20.6 (106.7) | -69.6 (206.7) | -13.1 (84.5) | -13.0 (123.2)
  Week 32: number analyzed (Participants) | 41 | 41 | 41 | 41
  Week 32 | -14.3 (106.3) | -75.8 (225.7) | -10.4 (93.0) | -20.9 (168.1)
  Week 40: number analyzed (Participants) | 40 | 41 | 39 | 43
  Week 40 | -24.8 (103.3) | -68.6 (211.0) | -26.9 (83.0) | -46.9 (138.0)
  Week 48: number analyzed (Participants) | 35 | 40 | 35 | 41
  Week 48 | -37.0 (132.7) | -82.4 (243.7) | -15.5 (83.2) | -41.2 (120.0)

35. Secondary Outcome: Mean Change From Baseline in CD19/Lymphocytes
Description: CD19/Lymphocytes was measured in percentages (%).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of CD19 per Leukocytes
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of CD19 per Leukocytes
  Week 2: number analyzed (Participants) | 38 | 40 | 42 | 40
  Week 2 | -0.3 (2.1) | -0.1 (3.0) | 1.0 (3.5) | 1.5 (5.9)
  Week 4: number analyzed (Participants) | 39 | 40 | 40 | 39
  Week 4 | 0.0 (2.9) | -0.5 (3.7) | 0.7 (3.3) | 2.8 (5.7)
  Week 8: number analyzed (Participants) | 38 | 40 | 39 | 40
  Week 8 | 0.1 (2.8) | -0.5 (4.2) | 0.7 (2.5) | 0.4 (6.4)
  Week 12: number analyzed (Participants) | 41 | 41 | 40 | 40
  Week 12 | -0.2 (3.2) | -1.0 (3.9) | -0.4 (3.1) | 1.7 (7.9)
  Week 16: number analyzed (Participants) | 38 | 42 | 38 | 42
  Week 16 | 0.0 (4.7) | -1.2 (5.0) | -0.4 (3.3) | 0.7 (5.9)
  Week 20: number analyzed (Participants) | 40 | 40 | 39 | 42
  Week 20 | -0.4 (3.8) | -2.1 (6.2) | -0.3 (3.0) | -0.2 (6.9)
  Week 24: number analyzed (Participants) | 39 | 39 | 42 | 43
  Week 24 | -0.9 (4.5) | -2.0 (6.5) | -0.6 (3.3) | -0.3 (7.3)
  Week 28: number analyzed (Participants) | 41 | 40 | 39 | 38
  Week 28 | -1.2 (5.4) | -2.5 (5.9) | -1.1 (3.3) | -1.0 (6.6)
  Week 32: number analyzed (Participants) | 41 | 41 | 41 | 41
  Week 32 | -0.4 (4.7) | -2.4 (5.5) | -0.6 (4.4) | -1.6 (6.3)
  Week 40: number analyzed (Participants) | 40 | 41 | 39 | 43
  Week 40 | -1.2 (4.7) | -2.6 (5.4) | -1.9 (4.2) | -3.4 (6.7)
  Week 48: number analyzed (Participants) | 35 | 40 | 35 | 41
  Week 48 | -1.2 (6.8) | -2.6 (7.2) | -1.6 (4.9) | -3.3 (6.2)

36. Secondary Outcome: Mean Change From Baseline in Aspartate Aminotransferase
Description: Aspartate Aminotransferase was measured in units per liter (U/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
U/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | -0.5 (8.8) | 0.2 (8.0) | 4.3 (43.1) | 0.0 (7.2)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.1 (11.2) | 0.2 (7.4) | -1.1 (7.6) | -1.9 (8.0)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -0.1 (8.7) | -1.5 (6.2) | 0.5 (13.0) | -1.1 (8.1)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 5.1 (27.0) | 0.9 (6.2) | -1.8 (10.0) | -2.9 (7.1)
  Week 16: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 16 | 0.4 (7.7) | 0.0 (6.3) | -2.3 (11.6) | -2.8 (8.4)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 44
  Week 20 | 4.1 (24.1) | 1.0 (11.5) | -0.7 (13.8) | -3.8 (8.1)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 0.6 (11.8) | 1.6 (10.4) | -1.8 (11.5) | -3.8 (8.4)
  Week 28: number analyzed (Participants) | 43 | 42 | 40 | 42
  Week 28 | 0.0 (12.3) | 0.0 (10.2) | -1.5 (11.1) | -3.4 (9.1)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 44
  Week 32 | -0.3 (11.0) | 0.3 (6.8) | -0.7 (12.9) | -3.4 (9.2)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -0.6 (10.2) | 0.1 (9.1) | -0.3 (11.5) | -1.5 (9.8)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 1.1 (10.8) | 0.1 (13.1) | 1.4 (13.4) | -2.1 (8.6)

37. Secondary Outcome: Mean Change From Baseline in Alanine Aminotransferase
Description: Alanine Aminotransferase was measured in units per liter (U/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
U/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | 2.4 (14.1) | 2.6 (10.6) | 0.5 (11.1) | -0.1 (8.6)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.8 (9.9) | -0.5 (8.5) | 0.9 (7.4) | 0.3 (8.2)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 0.2 (10.2) | -0.8 (8.3) | 5.3 (28.8) | -0.6 (9.6)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 7.0 (21.3) | 0.8 (14.3) | -0.8 (8.1) | -0.1 (7.6)
  Week 16: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 16 | 1.5 (13.3) | -0.4 (9.3) | 0.0 (10.3) | -1.1 (7.8)
  Week 20: number analyzed (Participants) | 43 | 43 | 42 | 44
  Week 20 | 5.3 (23.6) | -0.2 (10.2) | 1.4 (10.8) | -3.7 (6.3)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 3.1 (20.9) | 0.5 (14.1) | 2.0 (12.0) | -2.8 (7.7)
  Week 28: number analyzed (Participants) | 43 | 42 | 40 | 42
  Week 28 | 1.0 (13.9) | 0.7 (10.5) | -0.4 (9.3) | -2.7 (7.2)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 44
  Week 32 | 1.2 (13.4) | -0.5 (10.3) | 1.3 (10.8) | -3.2 (6.1)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -0.5 (13.4) | 2.6 (12.8) | 3.0 (12.9) | -0.7 (8.3)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 0.4 (11.5) | -1.2 (10.4) | 3.5 (17.0) | -1.1 (7.8)

38. Secondary Outcome: Mean Change From Baseline in Alkaline Phosphatase
Description: Alkaline Phosphatase was measured in units per liter (U/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
U/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | 1.8 (10.7) | 2.4 (10.6) | 1.5 (8.0) | -3.6 (10.1)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -1.7 (9.7) | 0.7 (9.2) | -0.7 (8.4) | -4.7 (9.4)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 1.7 (12.9) | 2.4 (12.7) | 1.8 (15.6) | -6.1 (11.0)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 2.2 (11.6) | 4.2 (16.4) | 1.9 (12.9) | -4.4 (11.8)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 3.1 (10.7) | 2.7 (13.0) | 0.0 (10.4) | -6.7 (12.8)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | 3.9 (14.0) | 1.4 (11.8) | 1.4 (11.8) | -7.4 (11.2)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 4.7 (15.0) | 3.7 (14.0) | 2.8 (11.6) | -2.7 (14.0)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | 2.8 (14.0) | 3.1 (14.2) | 1.9 (9.5) | -2.1 (13.5)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 3.8 (14.6) | 2.7 (16.0) | 3.2 (12.1) | 1.0 (15.9)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 2.4 (17.1) | 1.3 (13.1) | 2.7 (13.0) | -3.0 (18.0)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 2.6 (13.3) | 4.0 (16.8) | 5.5 (12.8) | -4.5 (18.8)

39. Secondary Outcome: Mean Change From Baseline in Gamma Glutamyl Transferase
Description: Gamma Glutamyl Transferase was measured in units per liter (U/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
U/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | 0.3 (7.6) | 2.0 (11.5) | 8.8 (68.9) | -3.4 (24.3)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 2.1 (8.7) | -1.3 (8.8) | 2.7 (28.5) | -6.5 (35.5)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 3.5 (23.0) | 0.3 (10.5) | -2.8 (49.3) | -9.2 (43.3)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 4.1 (21.0) | 0.5 (13.4) | -5.1 (29.3) | -8.3 (46.1)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 6.5 (20.2) | 2.1 (12.5) | -6.1 (45.0) | -10.6 (47.7)
  Week 20: number analyzed (Participants) | 43 | 44 | 42 | 44
  Week 20 | 3.5 (14.1) | 0.2 (13.4) | -3.7 (50.3) | -8.5 (50.5)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 7.1 (22.0) | 4.0 (18.7) | -0.4 (53.1) | -9.5 (47.2)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | 4.6 (25.7) | 2.2 (18.3) | -7.0 (46.8) | 0.0 (23.1)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 4.4 (28.6) | 1.5 (16.7) | -5.9 (44.5) | -8.2 (37.4)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 3.4 (41.3) | 5.7 (32.4) | 0.4 (10.1) | -9.1 (45.3)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 1.8 (11.4) | 5.3 (23.9) | 4.7 (21.6) | -9.8 (44.5)

40. Secondary Outcome: Mean Change From Baseline in Bilirubin
Description: Bilirubin was measured in micromols per liter (µmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
μmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | 0.35 (2.72) | -0.48 (2.71) | 0.28 (2.38) | -0.78 (3.13)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.07 (2.50) | -0.18 (2.09) | -0.05 (2.14) | -0.79 (2.80)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -0.09 (2.66) | -0.69 (2.22) | -0.19 (2.13) | -0.23 (2.80)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.04 (2.60) | -0.70 (2.74) | 0.37 (2.17) | -0.33 (3.28)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 0.06 (2.41) | -0.45 (2.43) | -0.20 (2.71) | -0.51 (3.64)
  Week 20: number analyzed (Participants) | 43 | 43 | 42 | 44
  Week 20 | -0.54 (2.89) | -0.38 (2.51) | 0.51 (2.81) | -0.30 (3.03)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 0.08 (2.75) | -0.14 (2.86) | 0.54 (2.18) | -0.38 (3.57)
  Week 28: number analyzed (Participants) | 43 | 42 | 40 | 42
  Week 28 | -0.10 (2.98) | -0.26 (3.23) | 0.79 (2.71) | -0.82 (2.61)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 44
  Week 32 | 0.09 (2.75) | -0.38 (2.61) | 0.93 (3.18) | -0.38 (3.61)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -0.26 (3.70) | 0.07 (3.18) | 1.03 (2.35) | -0.15 (2.64)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 0.69 (3.57) | -0.50 (3.12) | 0.79 (3.04) | -0.20 (2.52)

41. Secondary Outcome: Mean Change From Baseline in Direct Bilirubin
Description: Direct Bilirubin was measured in micromols per liter (µmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
μmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | 0.03 (0.92) | -0.06 (0.92) | 0.09 (1.12) | -0.24 (1.10)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.10 (1.03) | 0.03 (0.75) | -0.04 (0.82) | -0.10 (0.93)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 0.03 (0.91) | -0.18 (0.55) | -0.17 (0.86) | 0.03 (1.10)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 0.15 (0.99) | -0.07 (0.95) | -0.01 (1.06) | -0.05 (1.30)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 0.18 (0.81) | -0.01 (0.66) | -0.07 (1.04) | -0.01 (1.40)
  Week 20: number analyzed (Participants) | 43 | 43 | 42 | 44
  Week 20 | -0.04 (0.95) | 0.07 (0.91) | 0.02 (0.94) | 0.00 (1.19)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 0.05 (1.10) | 0.14 (0.95) | 0.08 (1.02) | -0.08 (1.25)
  Week 28: number analyzed (Participants) | 43 | 42 | 40 | 42
  Week 28 | 0.06 (1.06) | -0.06 (1.00) | 0.11 (0.80) | -0.06 (1.15)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 44
  Week 32 | 0.12 (1.16) | 0.05 (0.90) | 0.21 (1.21) | -0.04 (1.36)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 0.07 (1.31) | 0.03 (0.76) | 0.23 (1.00) | 0.07 (1.05)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 0.31 (1.34) | -0.05 (1.01) | 0.20 (1.25) | 0.08 (0.98)

42. Secondary Outcome: Mean Change From Baseline in Lactate Dehydrogenase
Description: Lactate Dehydrogenase was measured in units per liter (U/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
U/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | -3.3 (27.8) | -7.8 (21.2) | -5.9 (35.2) | -12.8 (24.8)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -3.0 (23.4) | -3.7 (37.0) | -5.6 (35.6) | -18.5 (34.1)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -5.7 (27.4) | -11.8 (31.5) | -9.2 (39.0) | -20.4 (37.4)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 3.0 (28.7) | -7.4 (34.6) | -11.1 (45.1) | -24.4 (39.0)
  Week 16: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 16 | -2.2 (25.5) | -11.1 (29.9) | -10.6 (48.6) | -22.4 (43.3)
  Week 20: number analyzed (Participants) | 43 | 45 | 41 | 44
  Week 20 | -0.7 (33.9) | -10.8 (37.0) | -9.9 (47.8) | -28.5 (32.1)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -4.5 (31.3) | -14.3 (31.5) | -14.6 (34.4) | -29.3 (32.2)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | 0.0 (40.8) | -16.0 (40.9) | -13.2 (35.0) | -34.8 (36.9)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 5.0 (55.0) | -9.9 (43.4) | -8.1 (33.5) | -22.9 (40.6)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -1.6 (38.1) | -2.9 (41.1) | -8.0 (28.4) | -20.5 (40.1)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -8.8 (35.2) | -4.2 (54.3) | -1.5 (32.7) | -16.0 (36.3)

43. Secondary Outcome: Mean Change From Baseline in Creatinine
Description: Creatinine was measured in micromols per liter (µmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
μmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | 0.9 (9.1) | -0.1 (8.0) | 1.5 (5.8) | 0.6 (7.2)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.8 (8.9) | -0.2 (9.3) | -0.6 (7.3) | -1.4 (8.2)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 0.5 (7.0) | 0.3 (7.6) | -0.5 (6.9) | 0.1 (8.4)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.3 (7.0) | 1.4 (7.5) | -0.4 (6.4) | -0.7 (8.2)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | -0.1 (9.8) | 1.0 (8.2) | 0.7 (6.8) | -1.1 (9.4)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | 0.7 (8.6) | 1.4 (10.2) | 0.8 (6.9) | -0.3 (7.7)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 0.0 (8.8) | 0.8 (8.8) | 0.3 (6.6) | 0.9 (9.7)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | 2.5 (10.0) | 2.7 (10.0) | 1.0 (7.8) | -0.9 (7.8)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 5.5 (35.7) | 0.5 (8.1) | 3.6 (7.8) | 1.6 (11.2)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 2.3 (9.5) | 2.2 (8.5) | 3.9 (6.0) | 3.0 (8.4)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 1.9 (10.6) | 0.7 (7.6) | 2.5 (5.2) | 2.9 (9.8)

44. Secondary Outcome: Mean Change From Baseline in Urea Nitrogen
Description: Urea Nitrogen was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | 0.28 (1.55) | -0.09 (1.23) | -0.05 (1.32) | -0.02 (1.31)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.07 (1.21) | -0.33 (1.52) | -0.14 (1.20) | 0.04 (1.19)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 0.06 (1.25) | -0.26 (1.22) | -0.19 (1.07) | 0.17 (1.59)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 0.03 (1.13) | -0.39 (1.31) | -0.29 (1.17) | -0.22 (1.15)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 0.19 (1.35) | -0.18 (1.40) | 0.19 (1.49) | -0.03 (1.41)
  Week 20: number analyzed (Participants) | 43 | 44 | 42 | 44
  Week 20 | -0.18 (1.29) | -0.20 (1.33) | -0.25 (1.22) | -0.16 (1.08)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | 0.08 (1.69) | -0.44 (1.38) | -0.13 (1.18) | -0.09 (1.50)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | 0.13 (1.38) | 0.03 (1.61) | -0.23 (1.26) | -0.22 (1.14)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 0.40 (2.37) | -0.30 (1.65) | 0.21 (1.17) | 0.10 (1.43)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 0.29 (1.54) | 0.10 (1.73) | 0.21 (1.20) | 0.14 (1.43)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 0.05 (1.22) | -0.31 (1.54) | 0.23 (1.38) | -0.02 (1.56)

45. Secondary Outcome: Mean Change From Baseline in Sodium
Description: Sodium was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | -0.1 (1.9) | -0.4 (2.4) | 0.1 (1.6) | 0.0 (2.2)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.3 (2.0) | -0.6 (2.1) | 0.3 (2.1) | -0.1 (2.4)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 0.1 (2.2) | -0.4 (2.4) | 0.3 (2.2) | 0.1 (2.3)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.3 (2.0) | -0.5 (2.0) | 0.2 (2.0) | 0.1 (2.3)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | -0.4 (2.3) | -0.2 (1.9) | 0.0 (2.0) | -0.2 (2.3)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | 0.3 (2.2) | -0.8 (2.2) | -0.1 (2.0) | -0.5 (2.4)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.1 (2.5) | -0.4 (2.2) | 0.0 (2.2) | -0.3 (2.1)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | 0.0 (1.9) | -0.4 (2.4) | 0.2 (1.9) | 0.1 (2.3)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 0.0 (2.3) | -0.8 (3.2) | 0.1 (2.1) | 0.2 (2.2)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -0.1 (2.2) | -1.2 (2.2) | -0.1 (1.6) | -0.3 (2.4)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.4 (2.0) | -1.1 (2.6) | -0.5 (1.7) | 0.2 (2.3)

46. Secondary Outcome: Mean Change From Baseline in Potassium
Description: Potassium was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 44 | 44
  Week 2 | 0.04 (0.45) | 0.15 (0.40) | 0.00 (0.36) | -0.03 (0.37)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.06 (0.44) | 0.08 (0.35) | -0.07 (0.41) | -0.12 (0.40)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -0.04 (0.40) | 0.11 (0.38) | 0.00 (0.35) | -0.07 (0.40)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | -0.01 (0.33) | 0.02 (0.31) | -0.07 (0.41) | -0.12 (0.34)
  Week 16: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 16 | -0.01 (0.34) | 0.16 (0.33) | -0.09 (0.42) | -0.05 (0.33)
  Week 20: number analyzed (Participants) | 43 | 45 | 40 | 43
  Week 20 | 0.04 (0.38) | 0.14 (0.33) | -0.04 (0.46) | -0.08 (0.37)
  Week 24: number analyzed (Participants) | 42 | 43 | 43 | 43
  Week 24 | 0.06 (0.43) | 0.07 (0.39) | 0.03 (0.33) | -0.11 (0.37)
  Week 28: number analyzed (Participants) | 41 | 43 | 40 | 43
  Week 28 | 0.09 (0.43) | 0.12 (0.47) | 0.06 (0.42) | 0.03 (0.45)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 0.03 (0.44) | 0.07 (0.44) | 0.10 (0.46) | -0.05 (0.38)
  Week 40: number analyzed (Participants) | 42 | 41 | 41 | 44
  Week 40 | 0.06 (0.33) | 0.16 (0.51) | 0.16 (0.39) | -0.06 (0.37)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.01 (0.30) | 0.00 (0.30) | -0.02 (0.39) | -0.07 (0.40)

47. Secondary Outcome: Mean Change From Baseline in Calcium
Description: Calcium was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | 0.008 (0.104) | -0.001 (0.103) | 0.004 (0.088) | -0.008 (0.092)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.007 (0.108) | -0.018 (0.099) | -0.018 (0.090) | -0.001 (0.086)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -0.006 (0.093) | -0.033 (0.117) | -0.014 (0.106) | -0.003 (0.089)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | 0.006 (0.108) | -0.011 (0.121) | -0.013 (0.097) | -0.004 (0.111)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | -0.025 (0.106) | -0.004 (0.088) | -0.013 (0.095) | -0.024 (0.119)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | -0.036 (0.116) | -0.020 (0.084) | -0.015 (0.108) | 0.005 (0.080)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.027 (0.106) | -0.026 (0.094) | -0.012 (0.095) | 0.007 (0.100)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | -0.031 (0.121) | -0.039 (0.091) | -0.016 (0.113) | -0.014 (0.092)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 0.003 (0.098) | -0.043 (0.099) | 0.019 (0.107) | -0.001 (0.105)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -0.027 (0.114) | -0.022 (0.115) | 0.006 (0.115) | -0.012 (0.105)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.013 (0.096) | -0.037 (0.119) | -0.004 (0.104) | -0.017 (0.110)

48. Secondary Outcome: Mean Change From Baseline in Phosphate
Description: Phosphate was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 44 | 43
  Week 2 | 0.044 (0.163) | 0.032 (0.192) | -0.047 (0.230) | 0.033 (0.168)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.004 (0.162) | -0.029 (0.185) | -0.070 (0.187) | 0.020 (0.163)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 0.006 (0.178) | -0.063 (0.225) | -0.028 (0.207) | 0.051 (0.187)
  Week 12: number analyzed (Participants) | 44 | 44 | 44 | 44
  Week 12 | 0.029 (0.159) | -0.004 (0.149) | -0.015 (0.236) | 0.045 (0.183)
  Week 16: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 16 | -0.010 (0.186) | 0.012 (0.182) | -0.025 (0.195) | 0.005 (0.178)
  Week 20: number analyzed (Participants) | 43 | 43 | 41 | 43
  Week 20 | -0.030 (0.208) | -0.037 (0.244) | -0.031 (0.177) | 0.013 (0.187)
  Week 24: number analyzed (Participants) | 42 | 43 | 43 | 43
  Week 24 | -0.013 (0.181) | -0.042 (0.160) | -0.040 (0.229) | 0.035 (0.200)
  Week 28: number analyzed (Participants) | 41 | 42 | 40 | 42
  Week 28 | -0.024 (0.189) | 0.008 (0.238) | -0.031 (0.232) | 0.037 (0.184)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 44
  Week 32 | -0.002 (0.217) | -0.056 (0.223) | 0.015 (0.220) | 0.030 (0.190)
  Week 40: number analyzed (Participants) | 42 | 41 | 41 | 44
  Week 40 | 0.018 (0.207) | 0.009 (0.196) | -0.022 (0.208) | 0.034 (0.224)
  Week 48: number analyzed (Participants) | 38 | 41 | 40 | 43
  Week 48 | 0.032 (0.183) | -0.012 (0.167) | -0.044 (0.214) | 0.035 (0.190)

49. Secondary Outcome: Mean Change From Baseline in Cholesterol
Description: Cholesterol was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | 0.00 (0.49) | -0.07 (0.46) | -0.06 (0.51) | -0.19 (0.47)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.08 (0.49) | -0.03 (0.46) | -0.07 (0.68) | -0.07 (0.57)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -0.09 (0.57) | -0.07 (0.46) | -0.15 (0.81) | -0.17 (0.59)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.14 (0.72) | -0.16 (0.61) | -0.23 (0.68) | -0.10 (0.75)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | -0.16 (0.80) | -0.16 (0.66) | -0.35 (0.80) | -0.27 (0.72)
  Week 20: number analyzed (Participants) | 43 | 44 | 42 | 44
  Week 20 | -0.27 (0.77) | -0.22 (0.60) | -0.42 (0.81) | -0.23 (0.85)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.12 (0.87) | -0.17 (0.66) | -0.28 (0.96) | -0.16 (0.78)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | -0.17 (0.89) | -0.37 (0.63) | -0.35 (0.97) | -0.29 (0.80)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | -0.13 (0.86) | -0.22 (0.63) | -0.16 (0.83) | -0.15 (0.81)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -0.34 (0.87) | -0.25 (0.80) | -0.19 (0.77) | -0.13 (1.15)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.40 (0.80) | -0.36 (0.74) | -0.23 (0.97) | -0.18 (1.09)

50. Secondary Outcome: Mean Change From Baseline in Triglycerides
Description: Triglycerides was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | -0.176 (1.593) | 0.046 (0.683) | 0.110 (0.855) | 0.183 (0.751)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.189 (1.212) | -0.004 (0.510) | -0.030 (0.471) | 0.084 (0.529)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -0.182 (1.554) | 0.076 (0.582) | -0.084 (0.498) | 0.046 (0.585)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.265 (1.445) | 0.088 (0.713) | 0.063 (0.578) | 0.009 (0.514)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | -0.164 (1.345) | 0.099 (1.488) | 0.142 (0.580) | 0.112 (1.035)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | -0.233 (1.391) | -0.104 (0.837) | 0.008 (0.622) | -0.060 (0.707)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.263 (1.515) | -0.045 (0.774) | -0.013 (0.608) | -0.030 (0.707)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | -0.013 (1.559) | -0.125 (0.782) | -0.043 (0.423) | -0.036 (0.663)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | -0.260 (1.418) | 0.045 (0.717) | 0.057 (0.532) | 0.112 (0.718)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -0.134 (1.175) | -0.159 (0.765) | 0.177 (0.821) | 0.022 (0.644)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.242 (1.516) | -0.149 (0.758) | 0.114 (0.507) | 0.054 (0.752)

51. Secondary Outcome: Mean Change From Baseline in Protein
Description: Protein was measured in grams per liter (g/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
g/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | -0.2 (3.7) | -1.2 (4.0) | -1.0 (4.2) | -1.1 (3.8)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -1.5 (4.4) | -1.6 (4.2) | -1.5 (4.7) | -1.7 (4.4)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -1.1 (4.4) | -2.1 (4.1) | -1.8 (5.7) | -2.0 (3.9)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.8 (3.8) | -1.3 (4.7) | -1.4 (5.2) | -1.2 (5.8)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | -1.2 (5.2) | -0.3 (4.1) | -2.3 (5.6) | -3.8 (5.0)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | -2.7 (6.0) | -1.6 (4.6) | -2.6 (4.7) | -3.1 (5.4)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -2.2 (7.5) | -1.8 (4.6) | -1.8 (5.5) | -2.0 (4.7)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | -3.1 (7.4) | -2.4 (4.6) | -2.5 (5.7) | -3.6 (6.4)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | -1.4 (6.9) | -1.5 (5.7) | -0.8 (5.0) | -1.9 (6.4)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | -2.2 (6.5) | -0.9 (5.0) | -1.8 (5.3) | -2.6 (6.1)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -2.3 (6.2) | -2.4 (5.9) | -0.9 (5.1) | -3.4 (6.4)

52. Secondary Outcome: Mean Change From Baseline in Albumin
Description: Albumin was measured in grams per liter (g/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
g/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | 0.1 (2.1) | -0.4 (2.4) | -0.5 (2.4) | -0.5 (1.9)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -0.5 (2.4) | -0.4 (2.3) | -0.2 (2.4) | -0.3 (1.9)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -0.3 (2.3) | -0.3 (2.5) | -0.3 (3.0) | 0.1 (2.2)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.1 (2.2) | 0.2 (2.7) | 0.2 (2.7) | 0.7 (3.0)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 0.0 (2.5) | 1.0 (2.5) | 0.1 (2.9) | -0.2 (2.9)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | -0.7 (2.7) | 0.1 (2.7) | 0.4 (2.4) | 0.4 (2.2)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.1 (2.9) | 0.0 (2.1) | 0.4 (2.4) | 1.2 (2.7)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | -0.7 (3.0) | -0.4 (2.3) | 0.1 (2.9) | 0.1 (2.6)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 0.6 (2.8) | -0.1 (3.0) | 0.9 (3.2) | 0.7 (2.8)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 0.1 (2.8) | -0.1 (2.9) | 0.2 (2.6) | 0.3 (3.0)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 0.1 (2.8) | -0.7 (3.0) | 0.2 (3.0) | -0.8 (3.5)

53. Secondary Outcome: Mean Change From Baseline in Glucose
Description: Glucose was measured in millimoles per liter (mmol/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
mmol/L
  Week 2: number analyzed (Participants) | 42 | 45 | 44 | 43
  Week 2 | 0.18 (0.75) | 0.26 (0.70) | 0.09 (0.78) | 0.13 (1.28)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 0.04 (0.71) | 0.03 (0.70) | -0.04 (0.90) | 0.11 (1.10)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | 0.17 (0.66) | 0.12 (0.90) | 0.23 (0.95) | 0.12 (1.16)
  Week 12: number analyzed (Participants) | 44 | 44 | 43 | 44
  Week 12 | -0.08 (0.69) | 0.08 (0.66) | -0.13 (0.79) | -0.15 (0.99)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 0.11 (0.77) | 0.06 (0.63) | 0.16 (0.92) | -0.18 (1.47)
  Week 20: number analyzed (Participants) | 43 | 44 | 42 | 43
  Week 20 | 0.16 (0.85) | 0.20 (0.84) | 0.13 (0.83) | -0.08 (1.01)
  Week 24: number analyzed (Participants) | 42 | 43 | 43 | 43
  Week 24 | -0.07 (0.85) | 0.05 (0.49) | -0.09 (0.73) | -0.22 (1.06)
  Week 28: number analyzed (Participants) | 39 | 43 | 40 | 43
  Week 28 | 0.22 (1.01) | 0.09 (0.76) | -0.01 (0.74) | 0.07 (1.22)
  Week 32: number analyzed (Participants) | 44 | 44 | 42 | 45
  Week 32 | -0.04 (0.72) | -0.07 (0.63) | -0.08 (0.65) | 0.06 (1.10)
  Week 40: number analyzed (Participants) | 41 | 41 | 41 | 44
  Week 40 | -0.05 (0.62) | 0.08 (0.71) | -0.09 (0.68) | -0.08 (1.07)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.14 (0.78) | -0.11 (0.61) | -0.06 (0.64) | -0.14 (1.25)

54. Secondary Outcome: Mean Change From Baseline in Lipase, Pancreatic
Description: Lipase, Pancreatic was measured in units per liter (U/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
U/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 44
  Week 2 | -1.1 (10.5) | 2.2 (11.9) | 0.1 (9.2) | -0.2 (7.5)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | -2.1 (9.8) | 0.9 (9.1) | 0.1 (10.6) | -1.2 (10.0)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -3.1 (9.2) | 3.7 (11.8) | 2.0 (20.0) | -1.8 (10.3)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -0.5 (8.7) | 1.0 (11.1) | -0.7 (13.4) | -0.6 (9.6)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 0.4 (7.4) | 2.7 (8.4) | 0.5 (11.3) | -0.2 (11.8)
  Week 20: number analyzed (Participants) | 43 | 45 | 42 | 44
  Week 20 | -0.6 (10.4) | 2.1 (8.0) | -0.9 (9.0) | -1.7 (9.3)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -0.5 (11.0) | -0.1 (9.1) | -0.1 (8.1) | 1.2 (11.8)
  Week 28: number analyzed (Participants) | 43 | 43 | 40 | 43
  Week 28 | 1.6 (13.1) | 1.7 (10.5) | 0.5 (11.9) | 1.7 (14.1)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 1.1 (15.1) | 1.0 (11.0) | 1.2 (10.6) | 3.8 (21.6)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 1.2 (11.0) | 1.3 (7.0) | -0.3 (8.9) | 2.5 (8.9)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 1.4 (10.1) | 2.2 (10.0) | 0.3 (10.7) | 3.7 (10.2)

55. Secondary Outcome: Mean Change From Baseline in Creatine Kinase
Description: Creatine Kinase was measured in units per liter (U/L).
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
U/L
  Week 2: number analyzed (Participants) | 42 | 45 | 45 | 43
  Week 2 | -3.0 (67.1) | -2.2 (55.6) | -2.2 (18.2) | 0.1 (46.5)
  Week 4: number analyzed (Participants) | 44 | 44 | 43 | 46
  Week 4 | 29.6 (218.4) | -6.2 (54.8) | 3.2 (22.0) | -16.9 (56.5)
  Week 8: number analyzed (Participants) | 44 | 43 | 44 | 44
  Week 8 | -4.9 (56.9) | -8.5 (52.7) | -1.5 (23.6) | -4.6 (122.1)
  Week 12: number analyzed (Participants) | 44 | 44 | 45 | 44
  Week 12 | -6.3 (57.5) | -8.4 (85.8) | -3.0 (22.4) | -29.4 (80.7)
  Week 16: number analyzed (Participants) | 44 | 45 | 43 | 45
  Week 16 | 0.9 (59.4) | -11.5 (105.1) | -7.5 (22.2) | -23.2 (106.3)
  Week 20: number analyzed (Participants) | 43 | 43 | 42 | 44
  Week 20 | -8.2 (60.0) | 5.9 (149.1) | -3.5 (22.2) | -33.4 (95.3)
  Week 24: number analyzed (Participants) | 42 | 43 | 44 | 44
  Week 24 | -6.4 (48.6) | -5.4 (123.7) | -2.6 (27.4) | -27.7 (98.9)
  Week 28: number analyzed (Participants) | 43 | 42 | 40 | 43
  Week 28 | -1.5 (67.3) | -19.1 (131.5) | -0.7 (25.4) | -36.7 (103.8)
  Week 32: number analyzed (Participants) | 44 | 44 | 43 | 45
  Week 32 | 2.0 (67.0) | -10.0 (167.0) | 34.0 (222.1) | -24.2 (91.2)
  Week 40: number analyzed (Participants) | 42 | 42 | 41 | 44
  Week 40 | 9.9 (109.1) | -20.4 (131.4) | -2.7 (25.4) | -16.3 (106.4)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | 7.8 (67.3) | -20.4 (138.3) | -3.6 (25.5) | -33.4 (106.5)

56. Secondary Outcome: Mean Change From Baseline in pH
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
pH
  Week 2: number analyzed (Participants) | 43 | 43 | 44 | 43
  Week 2 | -0.01 (0.66) | 0.03 (0.62) | -0.07 (0.67) | 0.15 (0.78)
  Week 4: number analyzed (Participants) | 43 | 43 | 43 | 43
  Week 4 | 0.10 (0.77) | 0.15 (0.52) | 0.06 (0.72) | 0.16 (0.74)
  Week 8: number analyzed (Participants) | 42 | 44 | 44 | 42
  Week 8 | -0.12 (0.79) | 0.00 (0.62) | -0.08 (0.56) | -0.04 (0.65)
  Week 12: number analyzed (Participants) | 44 | 43 | 43 | 42
  Week 12 | 0.00 (0.81) | 0.15 (0.69) | 0.03 (0.79) | 0.20 (0.83)
  Week 16: number analyzed (Participants) | 44 | 45 | 39 | 45
  Week 16 | -0.02 (0.61) | 0.00 (0.51) | -0.09 (0.81) | 0.11 (0.69)
  Week 20: number analyzed (Participants) | 42 | 43 | 41 | 43
  Week 20 | -0.11 (0.75) | -0.01 (0.59) | 0.06 (0.58) | 0.07 (0.88)
  Week 24: number analyzed (Participants) | 43 | 42 | 44 | 42
  Week 24 | 0.03 (0.85) | -0.01 (0.46) | -0.11 (0.81) | 0.02 (0.81)
  Week 28: number analyzed (Participants) | 44 | 42 | 42 | 41
  Week 28 | -0.13 (0.84) | -0.06 (0.57) | -0.05 (0.73) | -0.01 (0.69)
  Week 32: number analyzed (Participants) | 44 | 44 | 42 | 43
  Week 32 | -0.02 (0.75) | -0.03 (0.55) | -0.18 (0.66) | 0.09 (0.86)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -0.14 (0.81) | 0.19 (0.66) | -0.21 (0.81) | -0.07 (0.62)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.11 (0.66) | 0.06 (0.73) | -0.11 (0.74) | -0.08 (0.72)

57. Secondary Outcome: Mean Change From Baseline in Erythrocytes (/HPF)
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of Erythrocytes per HPF
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of Erythrocytes per HPF
  Week 2: number analyzed (Participants) | 43 | 43 | 44 | 43
  Week 2 | -6.8 (53.7) | 0.1 (8.4) | 0.2 (2.4) | 0.9 (7.9)
  Week 4: number analyzed (Participants) | 43 | 43 | 43 | 43
  Week 4 | -8.7 (52.6) | -0.8 (4.1) | 1.4 (10.5) | -0.6 (3.2)
  Week 8: number analyzed (Participants) | 42 | 44 | 44 | 42
  Week 8 | -8.7 (53.5) | -0.3 (6.9) | 0.4 (6.1) | 0.0 (6.8)
  Week 12: number analyzed (Participants) | 44 | 43 | 43 | 42
  Week 12 | -8.6 (52.6) | 1.3 (17.4) | -0.4 (2.4) | 17.4 (118.5)
  Week 16: number analyzed (Participants) | 43 | 45 | 39 | 45
  Week 16 | -5.7 (48.0) | -1.3 (4.1) | -0.6 (2.6) | -0.5 (5.5)
  Week 20: number analyzed (Participants) | 42 | 43 | 41 | 43
  Week 20 | -7.7 (53.7) | -1.0 (3.5) | -0.1 (3.9) | -0.6 (4.4)
  Week 24: number analyzed (Participants) | 43 | 42 | 44 | 42
  Week 24 | -7.2 (53.5) | -1.2 (3.9) | -0.3 (2.3) | -0.9 (4.6)
  Week 28: number analyzed (Participants) | 44 | 42 | 42 | 41
  Week 28 | -7.6 (51.3) | -1.3 (4.2) | -0.7 (2.9) | 3.0 (16.9)
  Week 32: number analyzed (Participants) | 44 | 44 | 42 | 43
  Week 32 | -8.5 (52.5) | 4.9 (41.8) | 0.0 (3.9) | 0.1 (4.5)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -9.1 (53.2) | 3.5 (18.8) | -0.5 (3.5) | 0.4 (5.4)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -9.7 (56.3) | -0.4 (5.4) | 1.9 (15.5) | 0.1 (4.0)

58. Secondary Outcome: Mean Change From Baseline in Leukocytes (/HPF)
Time Frame: From Baseline (Week 1) to Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % of Leukocytes per HPF
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
Number analyzed (Participants) | 45 | 45 | 45 | 47
% of Leukocytes per HPF
  Week 2: number analyzed (Participants) | 43 | 43 | 44 | 43
  Week 2 | -0.1 (11.4) | -1.4 (8.1) | -0.8 (2.9) | 2.9 (13.7)
  Week 4: number analyzed (Participants) | 43 | 43 | 43 | 43
  Week 4 | -0.2 (9.0) | -0.6 (8.5) | -0.7 (4.5) | 3.0 (12.6)
  Week 8: number analyzed (Participants) | 42 | 44 | 44 | 42
  Week 8 | -1.2 (10.4) | 4.8 (29.3) | -0.3 (6.8) | 3.0 (14.4)
  Week 12: number analyzed (Participants) | 44 | 43 | 43 | 42
  Week 12 | -1.1 (11.3) | 4.4 (42.2) | -1.3 (4.2) | 2.7 (13.9)
  Week 16: number analyzed (Participants) | 43 | 45 | 39 | 45
  Week 16 | 0.1 (9.6) | -1.6 (12.5) | -0.2 (9.6) | 1.8 (12.9)
  Week 20: number analyzed (Participants) | 42 | 43 | 41 | 43
  Week 20 | -0.1 (10.1) | 3.7 (13.3) | 0.4 (9.8) | 1.7 (4.0)
  Week 24: number analyzed (Participants) | 43 | 42 | 44 | 42
  Week 24 | -1.0 (10.9) | 10.7 (52.1) | -0.7 (4.5) | 0.4 (4.5)
  Week 28: number analyzed (Participants) | 44 | 42 | 42 | 41
  Week 28 | -0.2 (9.6) | 2.4 (9.7) | -1.1 (4.4) | 2.0 (10.1)
  Week 32: number analyzed (Participants) | 44 | 44 | 42 | 43
  Week 32 | -0.6 (10.8) | -0.5 (13.5) | -1.0 (5.4) | 4.1 (15.7)
  Week 40: number analyzed (Participants) | 42 | 43 | 41 | 44
  Week 40 | -1.6 (10.4) | 2.2 (19.8) | 1.4 (7.7) | 6.8 (30.9)
  Week 48: number analyzed (Participants) | 38 | 42 | 40 | 43
  Week 48 | -0.3 (8.9) | 10.8 (71.9) | -1.0 (4.0) | 0.8 (5.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline (Week 1) until end of the study (Week 48)
Arm/Group | SOC + Placebo iv Q4W (SS) | SOC + DZP 6mg/kg iv Q4W (SS) | SOC + DZP 24mg/kg iv Q4W (SS) | SOC + DZP 45mg/kg iv Q4W (SS)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/45 | 0/47
Serious Adverse Events (participants affected / at risk) | 6/45 | 5/45 | 6/45 | 5/47
Other Adverse Events (participants affected / at risk) | 19/45 | 23/45 | 22/45 | 21/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC + Placebo iv Q4W (SS) (N=45) | SOC + DZP 6mg/kg iv Q4W (SS) (N=45) | SOC + DZP 24mg/kg iv Q4W (SS) (N=45) | SOC + DZP 45mg/kg iv Q4W (SS) (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anastomotic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC + Placebo iv Q4W (SS) (N=45) | SOC + DZP 6mg/kg iv Q4W (SS) (N=45) | SOC + DZP 24mg/kg iv Q4W (SS) (N=45) | SOC + DZP 45mg/kg iv Q4W (SS) (N=47)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 5 (6) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4) | 3 (3) | 5 (6)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 4 (6) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (3) | 4 (4) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 3 (5) | 1 (1) | 2 (2)
Hepatic enzyme increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 5 (13) | 4 (4) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT02804763/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT02804763/SAP_001.pdf